#### **Document Coversheet**

Study Title: PROMIS WOMAN Education Program : ImProving ceRvical Cancer preventiOn Methods Among Muslim Americans WOMEN

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 7/8/2023 |
| NCT Number: | NCT05862844 |
| IRB Number | HM20024502 |
| Coversheet created: | 9/19/2024 |



Date: Saturday, July 8, 2023 9:07:32 AM

HM20024502

ID: HM20024502

Print Close

View: SF - Study Identification

HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN

## Study Identification

- 1. \* Select the Principal Investigator: Vanessa Lavene Sheppard
- 2. \* Study Title:

PROMIS WOMAN Education Program : ImProving ceRvical cancer preventiOn methods among Muslim AmerIcans WOMEN

- 3. \* Is this a student or trainee project in which activities will be carried out by that individual under your supervision (for example, dissertation or degree-required projects):
- Yes
- <sup>8</sup>C

If this project involves more than one student / trainee investigator, identify the primary contact here and list all student / trainee investigators in the Personnel section. Also ensure all are listed as protocol editors if they need to be copied on IRB correspondence and have authority to make edits.

- 4. \* Student/Trainee Investigator:
  - Asmaa Namoos
- 5. \* Please select the primary department or center that this study is being conducted under: Massey Cancer Center
- 6. Select the VCU IRB numbers assigned to studies that are:
  - 1. Associated with this study
- 2. Research registries this study will utilize
- Previously submitted versions of this study (closed, withdrawn, auto-withdrawn studies)

7/8/23, 9:07 AM

Title ₽ HM20021579 Participation of Muslim Women in Cervical Cancer Screening and HPV Vaccination Tamas Gal

7. Select all individuals who are permitted to edit the IRB protocol and should be copied on communications (study staff will be entered later). These individuals will be referred to as protocol editors:

| Last Name | Last Name First Name E-Mail | | Phone | Mobile |
|---|---|---|---|---|
| Gal | Tamas | tsgal@vcu.edu | 8046282123 | |
| Kim | Sun Jung | sjkim2@vcu.edu | | |
| LaRose | Jessica | jlarose@vcu.edu | | |
| Namoos | Asmaa | namoosa@vcu.edu | | |
| Perera | Robert | rperera2@vcu.edu | 8048272037 | |
| Sheppard | Vanessa Lavene | vlbsheppard@vcu.edu | | |

8. \* Select one of the following that applies to the project (selection will branch to new pages):
Note: VCU IRB offers guidance for many types of studies, including secondary data analysis studies, internet research, registries, EFIC, HUD, and Emergency Use protocols.

See https://research.vcu.edu/human\_research/guidance.htm



Research Project or Clinical Investigation [\*most exempt, expedited, and full board research studies]

| 0 |
|---|

| Humanitarian Use of Device for Treatment or Diagnosis |
|-------------------------------------------------------|
| 0 |

| ဗ္ဗ |
|---------------------------------------------------|
| 3ST |
| Humanitarian Use of Device for Clinical Investiga |
| = |
| ၓ |
| ≝ |
| _ |
| ₽ |
| ക്ര |
| ₹ |
| ä |
| ₽ |
| ψ |
| Š |
| ⊆ |
| ≌ |
| ₽ |
| ä |
| Ĕ |
| ₹ |
| _ |
| ( |
| L |

| ug, Biologic or Device |
|------------------------|
| of Investigational Dru |
| Emergency Use of |

| Use) |
|--------------|
| eatment |
| duct for Tr |
| nal Pro |
| nvestigatior |
| 함 |
| Access |
| Expanded |
| : Use ( |
| Treatment |

| Grant Review |
|--------------------|
| . Administrative |
| enter or Institute |
| ob<br>C |

Request for Not Human Subject Research Determination (i.e. request a letter confirming that IRB review is not

HM20024502

ID: HM20024502

View: SF2 - Federal Regulations

## methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn

## Federal Regulations

| ۴. |
|-------------------------|
| ≥ |
| 2 |
| ≠ |
| Ś |
| $\overline{\mathbf{o}}$ |
| ĕ |
| ≠ |
| 10 |
| ⊒ |
| 0 |
| 9 |
| _ |
| ≍ |
| 문 |
| _ |
| Ø |
| 'n |
| 'n |
| Ø |
| this |
| s this |
| * Is this |
| s this |

FDA regulated research includes all clinical investigations involving a test article and a human subject(s) that has been submitted for approval to the FDA or may be submitted in the future.

- the study involves an IND/IDE, abbreviated IDE, IND/IDE exemption, HUD, expanded access, or is otherwise Check Yes if
- the study involves a test article being administered or dispensed to subjects NOT according to a clinicians' medical judgment but rather, per the study protocol, OR subject to 21 CFR 56,
  - the study does not involve a test article but intends to provide safety or efficacy data to the FDA.

Yes

8 N

HM20024502

ID: HM20024502

View: SF2 - IRB Panel Setup

## PROMIS WOMAN Education Program: ImProving ceRvical cancer prevention methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

## **IRB Panel Setup**

No or not applicable

View: SF2 - Review Setup HM20024502

ID: HM20024502

7/8/23, 9:07 AM

## methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn

### Review Setup

| 1. * Select which study type best describes the majority of the study. Your response will help determine which |
|---|
| IRB panel should review this. |



Bio-Medical Research





Social/Behavioral/Education (SBE) Research

2. \* Which option(s) best describe the way(s) this study's procedures will be conducted? (Select all that apply.) This information may be used by the IRB in triaging studies during an emergency.



In-person interactions / interventions with participants



Remote interactions / interventions with participants



Secondary data/specimen analyses with or without contact with study participants

3. \* Would it be possible to convert in-person activities in your study to remote if there is an approved contingency protocol?

Yes, could convert to remote activities

4. \* Does this study involve greater than minimal risk:





ŝ

5. \* Review type requested: (subject to IRB approval):





Expedited



6. \* Is this study initiated by a VCU investigator or a sponsor:



Sponsor or industry initiated

The IRB has determined that the selected types of anticipated individual and social benefit apply to this study

categories will appear blank until the IRB has made a determination. If a category is not checked, it does not The below information is read-only to investigators, and the categories are set by the IRB during review. All apply to this study. This information may be used by the IRB in triaging studies during an emergency situation.

Scientific benefit

Educational benefit for student/trainee investigators leading their own study

The following information applies to studies being reviewed by the VCU IRB.

The IRB has determined that the selected Exempt and/or Expedited categories apply to this study.

The below information is read-only to investigators, and the categories are set by the IRB during review. All categories will appear blank until the IRB has made a determination. If a category is not checked, it does not apply to this study or the study is being reviewed by an external IRB.

#### 7. For Expedited Studies:

Is research that will be performed on individual or group characteristics or behavior OR will Category Research Data Involves the collection of data from voice, video, digital, or image recordings made for research purposes. Collection

Category Behavioral

employ a survey, interview, oral history, focus group, program evaluation, human factors evaluation, or quality assurance methodologies.

HM20024502

View: SF2 - Initial Setup Complete

HM20024502

ID: HM20024502

7/8/23, 9:07 AM

PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

## Initial Setup Complete

Protocol Progress:

**■ INITIAL SETUP** 

© BACKGROUND, RATIONALE & GOALS
③ RESEARCH PLAN
④ CONSENT PLAN
⑤ RISKS, PRIVACY & CONFIDENTIALITY
⑥ POPULATIONS WITH SPECIAL CONSIDERATIONS
⑦ INSTITUTIONAL REQUIREMENTS
⑧ DOCUMENTS

Click Continue below to go to the next section

View: SF2 - Background, Rationale and Goals HM20024502

ID: HM20024502

## PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

## Background, Rationale and Goals

1. \* Describe the study's background and what is currently known from the scientific literature, including citations, or upload a citation list in document upload. Use lay language whenever possible

Significance

International and national data about cervical cancer and HPV infection.

caused by the Human Papillomavirus (HPV), a sexually transmitted virus.3 Cervical cancer has been described as the screening tests.4 Early detection has been proven to improve patients' survival rate, where the 5-year survival rate of cancer was only 17.6%.5 The National Cancer Institute's cancer trends progress report has shown that about 81% of cervical cancer in 2020 and 340 thousand dying worldwide. I In the USA, the number of new cervical cancer cases in women aged 21 to 65 had cervical cancer screening in 2018 in the United States 6 On the other hand, almost half of Cervical cancer is one of the most common cancers among females, with over 600 thousand women diagnosed with 2022 was estimated to be 14,100. In Virginia, the American Cancer Society reported 310 new cases. 2 Most cervical silent killer,' as preinvasive and early invasive cervical cancer is most likely asymptomatic and detected only during patients with localized lesions has been reported to be 90.9% while that of patients with advanced-stage cervical cancer cases are preventable. According to the World Health Organization, almost all cervical cancer cases are he women diagnosed with invasive cervical cancer have not undergone cervical cancer screening. 7 Scope of the problem in Virginia.

most cervical cancer (90%) caused by HPV infection.2, 8 There are about 200,000 Muslims in Virginia, mostly living in he Richmond and the Northern Virginia area, where Muslim women seek care in the late stages of cervical cancer.9 The number of new cervical cancer cases in 2022 was estimated to be 14,100 in the U.S. and 310 in Virginia, with Our preliminary work showed that Muslim women face socio-structural barriers and health system complexity that prevent them from being integrated into healthcare services.10 Cancer epidemiological data is lacking about this marginalized group, which makes it difficult to conduct cancer prevention disparities research. Community Profile.

projection was 2.6 million (0.8%) in 2010 and expected to be 6.2 million (1.7%) in 2030.14 Muslim population growth is community in the United States today. Virginia has the second-largest Muslim population in the U.S. by the percentage 50% of American Muslims are foreign-born 11 Racially, American Muslims are very diverse religious groups in the U.S. with no majority race, split as 25% Black, 24% White, 18% Arab, 18% Asian, 7% mixed race, and 5% Hispanic (Figure 1).12 In terms of origin, Middle Eastern Countries represent 41% of the entire Muslim community in the U.S.13 In the American Muslims' lives and identities. The social structure in Muslim communities is built on a historical cultural and A total of 3.5 million American Muslims live in the United States (U.S.), representing 1% of the total population. Over Richmond Area 15 The population density correlates with the availability of Mosques. There are 18 religious centers (Mosques) in Virginia, 8 of them in the Richmond area.16 The two main sects within Islam are Sunni and Shia. They of the population, with an estimated 2.7% 12 Much of that population is concentrated in Northern Virginia and in the religious framework, which promotes patriarchal structures in families and in the larger Muslim society. Males in the agree on most of the fundamental beliefs, rules, and practices of Islam 17 Religion plays an important role in most egarding clothes and customs to maintain moral and social status. Women must cover arms, legs, and hair in the based on immigration and a high fertility rate, making the Muslim community roughly as numerous as the Jewish amily control decisions of the female family members. Muslim Women must follow the Islam recommendations last two decades, the population growth trajectory of the American Muslim community has been doubling; the

Halal food stores and restaurants in the Richmond area 19 Similarly, to other religious communities, religious schools products, such as pork, and there are specific rules about the processing of meat products. Therefore, the availability of Halal food stores is important for the Muslim community. According to the Google search engine, there are over 20 presence of males who are not in the woman's family.18 The Muslim Culture prohibits alcohol, non-Halal animal are important for Muslims; Virginia has over 30 religious schools and academic centers.20

The structure and everyday life of Muslim families are controlled by religion and related customs. A study classifies Muslim families into five types.21 These include:

- are older generations who do not want to adapt to the changing world or innovation. They are very sensitive to gender · Conservative Muslims who live by the Sharia (Islam religious laws) recommend all issues in their lives. Usually, they nteraction in public places such as clinics, schools, and even family events.
  - New Age Muslims are more interested in new things and open to other religions. They believe in education equity between males and females. They are typical of the middle class.
- · Societal Conformists are more interested in social norms than in religious customs, and they typically belong to a low socioeconomic class.
- Practical Strivers are affiliated with the religion by birth but not very religious. They are driven by success and wealth and are open to different cultures. They are typically more educated and enjoy good socioeconomic status.
- · Liberals typically from the millennial age group, are not religious and are interested in traveling and exploring new communities and traditions. Identity and individuality are important to them.

orce changes on them. Changes in behavior can only originate from inside the community. This is why it's important to gender preference of healthcare providers, rejection of pork-based medical products (e.g., gelatin), difficulties making The cultural and religious background influences an individual's behaviors, attitudes, and beliefs toward health. Even ndependent decisions, as well as lack of education about diseases. These limitations might be the results of Islamic understand these cultural challenges. All these obstacles present difficulties to under-served Muslim women.18, 22 As mentioned above, the Muslim community is generally suspicious of outsiders, especially if those outsiders try to mention the objective and perceived barriers the Muslim community faces related to healthcare services, including cultural beliefs and practices. Other limitations may be due to suboptimal healthcare services provided by the U.S. hough this project focuses on how individual cultural and religious beliefs affect healthcare decisions, we have to mplement a Community-Based Participatory Research (CBPR) project to ensure that community leaders and nealthcare system due to the lack of cultural competency, such as the unavailability of female providers who members understand the research and advocate from the inside.

Cervical cancer disparities among Muslim women (Preliminary work).

complexity are some challenges that Muslim women encounter, leading to disparities in prevention rates 25 Preliminary adhere to their religion, they have difficulties finding suitable Health Care Providers (HCPs) in the U.S. and often do not work: Our prior research within a large academic health system revealed that nearly 65% of Muslim women diagnosed screening and HPV vaccination. To achieve this, a survey was conducted with 100 participants. The survey comprised about HPV infection, vaccination, cervical cancer risk, or screening programs, not to mention how these relate to each census data does not include religious affiliation.23 National statistics of cervical cancer incidence and mortality rates among Muslim women are lacking 24 Language barriers, transportation difficulties, and the U.S. healthcare system's other.10 Key barriers for Muslim women in the clinic were the language, the gender of the providers, and the medical sectional mixed-methods pilot study to narrow the gap in the literature and assess the sociocultural factors, religious authority interferes with certain medical services, such as gynecological exams.26 Since most Muslim women firmly seek care 10 Prior research has lacked a consistent unifying theoretical approach to framing how multiple factors at various validated scales, including demographics, religiosity, modesty measures, perceived religious discrimination, Muslim women in VA. The study used in-depth interviews and found that most participants had minimal information staff's lack of understanding of their cultural and religious customs 9 Islam is strict about women's behavior, and its prevention to reduce cancer-related morbidity and mortality.9 To address these disparities, we established a crossbeliefs, medical knowledge, and attitudes related to HPV vaccination uptake and cervical cancer screening among The American healthcare system provides very little epidemiological data about the Muslim community as the U.S. n the quantitative study, we investigated the factors that affect Muslim women's decision to seek cervical cancer different levels contribute to prevention and care reluctance. A better understanding of these factors and their with cervical cancer presented at late stages, which further reinforces the need to focus on promoting cancer interaction can guide novel, theory-based strategies to improve cervical cancer screening rates.

medical mistrust, health literacy screening, and primary care assessment survey trust. Additionally, the survey included questions on knowledge, attitude, and practice concerning cervical cancer prevention

naving heard of HPV were higher for respondents with higher education (OR=6.84; CI=1.42, 33.03) and lower for those hose with higher religiosity were less likely to have heard of it. The manuscript is currently under review. The odds of were more likely to be aware of HPV. Furthermore, education level and religiosity score were found to be significantly he pap smear test, and the awareness of HPV was generally low. Unmarried, educated women with higher incomes The results showed that although most Muslim women were aware of cervical cancer, very few had heard of or used associated with HPV awareness. Respondents with higher education were more likely to have heard of HPV, while with higher religiosity (OR=0.74, CI=0.57, 0.96).

Medical school curriculum and training program.

training for medical professionals. However, we found no published resources for teaching medical trainees about the developed using a framework adopted by the ACGME. The research team is created an effective cultural competency training session for second-year medical students prior to entering their clinical rotations. The session was one part of a month-long course at the University of Michigan Medical School. The integration of cultural competency training into a medical school's curriculum is essential to produce providers equipped to care for a diverse patient population. This The Liaison Committee on Medical Education and the ACGME have called for the integration of cultural competency Muslim Americans are a historically underrepresented and understudied population facing unique health disparities. care for Muslim patients. To address disparities in healthcare faced by Muslims, a cross-cultural training session for medical students was implemented by Sarsour et al. in 2021 for caring for Muslim patients 27 This session was session establishes a teaching model for how to train medical trainees to care for Muslim patients. Muslim community needs and cultural competency of the health system.

hat is culturally competent and sensitive to the unique beliefs and practices of Muslim patients. Some of the healthcare A systematic review found that meeting the healthcare needs of the Muslim community requires a healthcare system needs specific to the Muslim community may include 18:

- Modesty accommodations during medical exams and procedures: Muslim patients may have specific preferences egarding gender-specific care and modesty during medical exams.
- Accommodations for prayer and fasting during hospitalization. During certain times of the year, Muslims may fast from dawn until dusk, which may affect their medical treatment plan. Additionally, Muslims may need to pray multiple times a day, which may require specific accommodations during hospitalization.
- Halal food and medication options: Many Muslims follow dietary restrictions that require them to eat halal meat, which must be slaughtered and prepared according to specific religious guidelines.

Additionally, healthcare facilities should provide resources and accommodations to meet the specific needs of Muslim nealthcare environment that respects and accommodates the unique needs of the Muslim community can improve nealthcare providers. This training should include education on Muslim cultural beliefs, practices, and healthcare To address these needs, the healthcare system should prioritize cultural competency and sensitivity training for patients, such as private spaces for prayer, halal food options, and gender-specific care. Creating an inclusive needs, and provide opportunities for healthcare providers to learn from and work with Muslim communities. Muslim women and access of cervical cancer prevention support: No interventional program in VA nealth outcomes and promote health equity for all patients 28, 29.

depending on location and other factors. The only support they can get from their healthcare providers and clinics may offer culturally sensitive services that take into account the specific needs of Muslim women, such as providing female cause cervical cancer. There are various healthcare providers and clinics across the United States that offer cervical provide services to women regardless of their ability to pay and may offer language or cultural assistance to women women who are socially isolated such as Muslim women? Unfortunately, the literature review shows no intervention programs specifically tailored for Muslim women in the United States, as the availability of such programs may vary nealthcare providers or offering prayer accommodations. Muslim women can seek out these services by contacting cancer prevention programs, including Planned Parenthood and community health centers. These programs often regular screening every three years until age 65. The screening can be done through a Pap test, which checks for abnormal cells on the cervix, or an HPV test, which checks for the presence of the human papillomavirus that can who need it. Hereby, we ask important questions: are these programs fit for all women including the conservative The American Cancer Society recommends that women begin cervical cancer screening at age 21 and continue heir local health department or community organizations that serve their community.

educational material.33 A similar base to Padela et al.'s work but in a form of a focus group was tested in Scotland with a small population of Muslim women to promote colorectal, breast, and cervical cancer screening and demonstrated a nsurance status) and not cultural or religious considerations.30 To the best of our knowledge, no screening programs mprovement of perception of screening benefits and harms, albeit being statistically insignificant.32 A study by Wyatt The National Breast and Cervical Cancer Early Detection Program (NBCCEDP) was initiated in 1990, serving all U.S. previous 5 years for cervical cancer, this program only targets women based on their eligibility (i.e., age, income, and ates was built and assessed by Padela et al. in 2018 and demonstrated success in regard to immediate and delayed oopulation. An educational program intervention targeted to Muslim women to improve their breast cancer screening ikelihood of screening.31 Another intervention in the form of a video was tested by Pratt et al. with Somali American Although there are no specifically tailored interventions for promoting only cervical cancer screening for the Muslim and territories. Even though this program resulted in the screening of more than 600,000 women in the U.S. in the et al. tested educational brochures with a Muslim population in New York City and found a significant difference in oopulation, there are some already tested programs that included outcomes related to cervical cancer in this breast and cervical cancer knowledge, mammography, and pap smear screening as a result of providing the Muslim women to investigate its effect on participation in breast and cervical cancer screening and found an or campaigns were explicitly designed to be hospitable for Muslim women in the U.S. on national level. positive impact regarding knowledge and willingness to utilize screening services.34

n summary, hesitancy in cancer screening may explain, in part, the notable disparities in stage at diagnosis of cervical cancer observed among Muslim women. To date, the few studies aimed at determining factors contributing to the lack characteristics and cultures; thus, it is essential to understand how these factors contribute to the acceptance of the prevention and screening process. The sequential studies proposed herein aim at informing the science of cervical cultural, and systems-level factors contributing to disparities. Muslim women are characterized by a unique set of of cancer screening participation among Muslim women have not thoroughly investigated the social, behavioral, cancer prevention among Muslim women by using a theory-driven framework using a two-arms study design to mprove the cervical cancer disparities among Muslim women.

Community-Engaged Research Framework

Trust and mistrust play an important role in the Muslim community's social interactions, which face discrimination in the promote it. The Mosques are the centers of social interaction in Muslim communities. This project needs to engage the U.S. every day. This research will only be able to recruit participants if community leaders understand and actively mams at Mosques in and around Richmond, VA.

the cancer-related health and well-being of their communities. Our project has a 12-month planning period that focuses on building community capacity, developing community partnerships, and establishing community volunteers' networks, The community-engaged framework will implement a Community Action Model (CAM). The CAM is a five-step process sustainability plan. The CAM is fit for the community engagement part of our project due to the capability to involve the intending to advance health equity, and 2) Build the capacity of communities to create sustainable changes to improve community members in every aspect of the design, implementation, and evaluation of these community action plans. whose purpose will be to design community-driven strategies to eliminate cervical cancer disparities in the Muslim that starts with recruiting and building relationships with community partners and developing and implementing a community members to understand and command the policies, systems, and environment that affect their lives The CAM was selected to inform the CBPR approach due to the main aspects of the model that help 1) The community in the Richmond area,

cancer, screening for it, and HPV vaccination. The second step is community diagnosis; the research team will support community leaders in developing the research plan to outline their research questions and methodology to understand deliver their results back to community members. The fourth step is an action plan; the research team develops and implements a pilot or demonstration project that shows the chosen action/activity's feasibility and effectiveness. The ifth step is to build the capacity to maintain and enforce the action project teams by developing and implementing a between the research team and Imams of Mosques, and providing all information they need to understand cervical cervical cancer's local implications. The third step is the analysis and presenting findings; the research team must The first step of the CAM is recruiting and training community leaders inside Mosques, building the relationships sustainability plan.

Community-Engaged Infrastructure

The study will be based in Virginia, home to a diverse population of over 250,000 Muslims, most living in Northern and

Commonwealth University and the Islamic Center of Virginia (ICR) by establishing Community Advisory Boards (CABs) Central Virginia. The population density correlates with the availability of Mosques, ethnic food stores and restaurants, and Muslim schools. The project will work toward building a strong community partnership between the Virginia and engaging Community Peer Researchers (Figure 2).

suggested by previous studies. We will target scholars with expertise in behavioral interventions, Islamic theology, and aw, as well as community-based participatory research to include in the committee. The two main sects of Islam are participation in the study. Getting permission from Mosque leaders to be at the Mosque in person during worship day community members to influence research activities. The CABs will include religious leaders from the ICR, which is religious leaders as members of the CABs.35 Using religious voices to communicate about our project will enhance CABs commonly formalize the academic-community partnerships that guide CBPR by providing a mechanism for American women as possible 17 There are no female religious leaders in Mosques, so we can only have male Sunni and Shia, therefore we decided to recruit both Sunni and Shia representatives to reach as many Muslim (Friday) will greatly help with the study progress.

the quality of the service that is provided for its patients, and it also has a diverse set of researchers and research staff Community Partnerships: For this study, the Massey Cancer Center (MCC), Virginia Commonwealth University, will be partnering with the community. MCC is located in Richmond, VA, in our target geographic area. MCC is well-known for mproving healthcare services and cancer outcomes among minorities in the Richmond area, which fits well with the who are well-versed in community-involved research. One of the MCC goals is to reduce cancer disparities by goals of our project. The partnership with MCC will significantly enhance our research project as it will provide ecognition and trust. It will also secure better relationships with the community.

to their shared life experiences as women having the same religion and traditions and familiarity with social norms. The communicate with the research team. Our preference is to recruit women and peer researchers who have been visiting Most Islamic centers open on Fridays, and the is hours when which people practice their worships are usually between Mosque rules and etiquette. We will also pursue building a strong relationship with Muslim women who are coming to ake classes inside the Mosque. Peer researchers will develop a better connection with the research participants due esearchers to cover cultural sensitivities and reach a high number of Muslim women. Peer researchers will serve as dentified themselves as Muslims. Age plays an important role in Muslim culture; participants will be more trusting to peer researchers will have to be trained in research processes. Our expectation is that the targeted peer researcher 12-1 PM, during regular business hours in the U.S. To overcome this problem, we will have 2 peer researchers, and cohort will not have difficulties with training, but they might have challenges regarding the schedule and availability. advanced English skills (speak, write, and read) and use technology to easily overcome the language barriers and partners with full involvement and authority in research processes. The eligibility criteria will be adult women who the Mosque for at least 5 years to have enough experience with interacting with Mosque visitors and Islamic and Since we will not have the opportunity of having Muslim women in the CABs, we decided to engage female peer what more grown community members provide more than the new generation. Peer researchers should have each woman will cover a day per month.

#### References

- GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2021. 2. Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA: A Cancer Journal for Clinicians. 2021; 71:7-1. Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, et al. Global cancer statistics 2020:
- World Health Orgininzation WHO. Human papillomavirus (HPV) and cervical cancer. 2020.
- 4. Pandey D, Shetty J, Sambhaji C, Saxena PU, Mishra D, Chawla A. Cervical Cancer as a silent killer: A rare case report with review of literature. J Cancer Res Ther. 2015; 11:653.
  - 5. Howlader et al. Cancer statistics review, 1975–2012. National Cancer Institute, Bethesda. 2015, Available from: https://seer.cancer.gov/archive/csr/1975\_2012/.
    - National Cancer Institue. Cervical Cancer Screening. 2020.
- 7. Akers AY, Newmann SJ, Smith JS. Factors underlying disparities in cervical cancer incidence, screening, and freatment in the United States. Curr Probl Cancer. 2007; 31:157-81.
  - 8. Organization WH. Human papillomavirus (HPV) and cervical cancer. 2020 [12/31/2021]; Available from: https://www.who.int/news-room/fact-sheets/detail/human-papillomavirus-(hpv)-and-cervical-cancer.

9. Namoos A, Abosamak NE, Abdelkarim M, Ramadan R, Phillips B, Ramadan D, et al. Muslim Women and Disparities in Cancer Diagnosis: A Retrospective Study. Journal of Muslim Minority Affairs. 2021; 41:541-7

- 10. Namoos A, Sheppard V, Abdelkarim M, Abosamak N, Ramadan R, Gal T. Explore Cervical Cancer Prevention Methods among Conservative Muslim American Women in Virginia: An Exploratory Qualitative Study. Research
- Membership Study. Collected by the Association of Statisticians of American Religious Bodies (ASARB).," Association 11. Association of Statisticians of American Religious Bodies. "2010 US Religion Census: Religious Congregations & of Religion Data Archives, 2010.
- 12. World Population Review. Muslim Population by State 2022. 2022. [05/04/2022.]; Available from:
  - https://worldpopulationreview.com/state-rankings/muslim-population-by-state.
- 13. Pew Research Center. U.S. Muslims Concerned About Their Place in Society, but Continue to Believe in the American Dream. 2017. [05/04/2022.]; Available from: https://www.pewforum.org/wp
  - content/uploads/sites/7/2017/07/U.S.-MUSLIMS-FULL-REPORT-with-population-update-v2.pdf.
- Pew Research Center's Religion & Public Life Project. The Future of the Global Muslim Population. 2011. 05/04/2022]; Available from: www.pewforum.org/2011/01/27/the-future-of-the-global-muslim-population/.
- Virginia.: StatChat; 2021 [05/04/2022]; Available from: https://statchatva.org/2021/06/08/who-practices-what-religion-15. Sen S. Who Practices What Religion Where in Virginia? Weldon Cooper Center for Public Service, University of where-in-virginia/.
  - 16. Google Maps. Religious Centers in Virginia. 2021.
- 17. Sunnis and Shia: Islam's ancient schism.: BBC News.; 2016. [05/04/2022.]; Available from:
  - https://www.bbc.com/news/world-middle-east-16047709.
- 18. Attum B, Hafiz S, Malik A, Shamoon Z. Cultural Competence in the Care of Muslim Patients and Their Families. StatPearls. Treasure Island (FL)2021
- 19. Gooogle Maps. How many halal stores in Richmond area. 2021.
  - 20. Google Maps. Muslim schools in Virginia. 2021.
- 21. Rishi B. Islamic perspectives on marketing and consumer behavior : planning, implementation, and control. 2015.
  - 22. Martin MB. Perceived Discrimination of Muslims in Health Care. Journal of Muslim Mental Health. 2015; 9.
- 23. Laird LD, Amer MM, Barnett ED, Barnes LL. Muslim patients and health disparities in the UK and the US. Arch Dis Child, 2007; 92:922-6.
  - 24. Abboud S, De Penning E, Brawner BM, Menon U, Glanz K, Sommers MS. Cervical Cancer Screening Among Arab Women in the United States: An Integrative Review. Oncol Nurs Forum. 2017; 44:E20-E33.
    - 25. Tackett S, Young J, Putman S, Wiener C, Deruggiero K, Bayram J. Barriers to healthcare among Muslim women: A narrative review of the literature. Women's Studies International Forum. 2018; 69.
      - 26. Vahabi M, Lofters A. Muslim immigrant women's views on cervical cancer screening and HPV self-sampling in Ontario, Canada. BMC Public Health. 2016; 16:868.
- 27. Sarsour NY, Hammoud MM. Integration of Arab and Muslim Health Education Into a Medical School Curriculum.
- 28. Padela AI, Gunter K, Kilawi A. Meeting the healthcare needs of American Muslims: Challenges and strategies for nealthcare settings. Institute for Social Policy and Understanding: Institute for Social Policy and Understanding 2011 June 2011.
- 29. Padela AI, Gunter K, Killawi A, Heisler M. Religious Values and Healthcare Accommodations: Voices from the American Muslim Community. Journal of General Internal Medicine. 2012; 27:708-15.
  - 30. Centers for Disease Control and Prevention. About the National Breast and Cervical Cancer Early Detection
- Program. 2023; Available from: https://www.cdc.gov/cancer/nbccedp/about.htm. 31. Padela AI, Malik S, Ally SA, Quinn M, Hall S, Peek M. Reducing Muslim Mammography Disparities: Outcomes From a Religiously Tailored Mosque-Based Intervention. Health Education & Behavior. 2018, 45:1025-35.
- 32. Pratt R, Mohamed S, Dirie W, Ahmed N, Lee S, VanKeulen M, et al. Testing a Religiously Tailored Intervention with Somali American Muslim Women and Somali American Imams to Increase Participation in Breast and Cervical Cancer Screening. J Immigr Minor Health. 2020; 22:87-95.
  - 33. Wyatt LC, Chebli P, Patel S, Alam G, Naeem A, Maxwell AE, et al. A Culturally Adapted Breast and Cervical Cancer Screening Intervention Among Muslim Women in New York City: Results from the MARHABA Trial. Journal of Cancer Education. 2022; 38:682-90.

34. Christie-de Jong F, Kotzur M, Amiri R, Ling J, Mooney JD, Robb KA. Qualitative evaluation of a codesigned faithbased intervention for Muslim women in Scotland to encourage uptake of breast, colorectal and cervical cancer screening. BMJ Open. 2022; 12.

- 35. Elius M. Islamic View of Women Leadership as Head of the State: A Critical Analysis. Arts Faculty Journal.
- Framework in Communication Research: Exploring Parallel, Serial, and Moderated Mediation. Health Communication. 36. Jones CL, Jensen JD, Scherr CL, Brown NR, Christy K, Weaver J. The Health Belief Model as an Explanatory 2014; 30:566-76.
- 37. Chun Tie Y, Birks M, Francis K. Grounded theory research: A design framework for novice researchers. SAGE Open Medicine 2019, 7
- 39. Baruth M, Wilcox S, Laken M, Bopp M, Saunders R. Implementation of a Faith-Based Physical Activity Intervention: ntersection of Science and Practice to Improve Health Equity. American Journal of Public Health. 2010; 100:S40-S6. 38. Wallerstein N, Duran B. Community-Based Participatory Research Contributions to Intervention Research: The nsights from Church Health Directors. Journal of Community Health. 2008; 33:304-12.

# $2.\ ^*$ Describe the study hypothesis and/or research questions. Use lay language whenever possible.

Aim 1b. We will conduct individual interviews with key stakeholders in our Community Advisory Board (Muslim religious acceptance of cervical cancer screening and prevention. This aim includes the Phase III (Efficacy) of the ORBIT model. participants with the same eligibility criteria as in Aim 1, who have not participated in our previous studies, and conduct leaders (N=4)) to receive feedback on the developed materials and inform the intervention program. This aim includes a single-arm pilot trial. H2. We hypothesize that the religiously tailored and culturally appropriate intervention program H1. Participants will show significant improvements in knowledge and acceptance of cervical cancer prevention after Aim 2. We will test the preliminary efficacy of the religiously tailored and culturally appropriate intervention program. will be feasible to conduct as evidenced by meeting enrollment targets and the ability to implement the program as planned. H3. The intervention will be acceptable as evidenced by engagement (>60%) and retention (>80%), and Aim 3. We will test the feasibility and acceptability of the religiously tailored and culturally appropriate intervention the intervention. To test this hypothesis, we will conduct a pre-post survey to examine changes in knowledge and program which includes education and experiential practice/communication skills training. We will recruit 20 he Phase II (Preliminary Testing) of the ORBIT model (proof of concept, prepare the pilot) satisfaction survey ratings.

# 3. \* Describe the study's specific aims or goals. Use lay language whenever possible.

competency of healthcare providers related to the Muslim culture at the VCU health system. Our ongoing work with the methods. The secondary outcome is the acceptability and confidence/trust in cervical cancer prevention methods such and HPV-Vax. The Muslim Community Partners (MCPs) will collaborate with our institute (VCU) by reaching out to four Muslim community has informed us about the community's needs. In this project, we will implement an interventional motivator for Muslim families to change. The primary outcome is increasing awareness of cervical cancer prevention interventions, which combine health-related religious teachings and scientific information about the benefits of CC-S convince women to join our study, reach out to a high number of MAW, and because religious voices will be a good Islamic religious centers in Virginia. Partnership with Islamic centers is valuable to our project due to their: ability to program guided by a community-based participatory approach utilizing expert-led education sessions and peer-led Our team also investigates the barriers faced by MAW in the US healthcare system by evaluating the cultural

The research questions are: Would MAW intend to do cervical cancer screening and uptake the HPV Vaccination after an education program supported by the Mosques that they frequently visit?

The aims of the study are:

Aim 1b. We will conduct individual interviews with key stakeholders in our Community Advisory Board (Muslim religious leaders (N=4)) to receive feedback on the developed materials and inform the intervention program. This aim includes the Phase II (Preliminary Testing) of the ORBIT model (proof of concept, prepare the pilot).

acceptance of cervical cancer screening and prevention. This aim includes the Phase III (Efficacy) of the ORBIT model. participants with the same eligibility criteria as in Aim 1, who have not participated in our previous studies, and conduct a single-arm pilot trial. H2. We hypothesize that the religiously tailored and culturally appropriate intervention program H1. Participants will show significant improvements in knowledge and acceptance of cervical cancer prevention after Aim 2. We will test the preliminary efficacy of the religiously tailored and culturally appropriate intervention program. will be feasible to conduct as evidenced by meeting enrollment targets and the ability to implement the program as planned. H3. The intervention will be acceptable as evidenced by engagement (>60%) and retention (>80%), and the intervention. To test this hypothesis, we will conduct a pre-post survey to examine changes in knowledge and Aim 3. We will test the feasibility and acceptability of the religiously tailored and culturally appropriate interventior program which includes education and experiential practice/communication skills training. We will recruit 20 satisfaction survey ratings.

For these aims, we will use a survey that includes:

Pre-test survey, the scales are:

- Demographic
- 2. Perceived Discrimination
- Religious Discrimination
- Spiritual Health Locus of Control
  - 5. Modesty
- 6. Cervical Cancer Knowledge
  - 7. Perceived risk
- 8. Cuse of action 9. Self-efficacy
- 10. Attitude about CC screening
- 11. HPV vaccination acceptability

Prost-test survey, the scales are:

- 2. Perceived Discrimination
  - 3. Religious Discrimination
- 4. Spiritual Health Locus of Control.
  - 5 Modesty
- 6. Cervical Cancer Knowledge
  - 7. Perceived risk
- 8. Cuse of action
- 9. Attitude about CC screening
- 10. HPV vaccination acceptability
- 10. hr v vacciliation acceptability 11. General Self-Efficacy Scale (GSES)
- 12. Cervical Cancer Screening Self-Efficacy Scale

Satisfactory survey are:

- -Experience with the intervention.
  - Acceptability of content
- -Acceptability of delivery

## 4. \* Describe the scientific benefit or importance of the knowledge to be gained:

iterature shows the general lack of knowledge of Muslim women that are related to cervical cancer, there is a lack of educational intervention programs targeted toward Muslim women. Our study will implement the first educational program for Muslim women in the US, thus the effectiveness of educational programs in conservative communities The Muslim population represents a significant, and increasingly growing, portion of the US population. Although

## 5. \* Describe any potential for direct benefits to participants in this study:

The study will provide valuable information for the Muslim community or the general population, increase knowledge will increase the seeking for care: cervical cancer screening. Decreasing vaccine hesitancy

- 1. By the end of year one, 5% of the conservative Muslim Women in Richmond, Virginia will know that the HPV vaccine is safe and effective.
- 2. By the end of year one, 5% of conservative Muslim women in the Richmond Virginia Area will know that the HPV vaccination will not cause their children to become sexually active before marriage.
- 3. By the end of year two 8% of conservative parents of Muslim girls in the Richmond Virginia Area will know that the HPV vaccination does not impact fertility and will permit administration of the vaccine to their daughters and sons
- By the end of the program most women will seek for Cervical cancer screening: pap smear test

## communities to respond to community-identified needs, or ways the study will strengthen the well-being of 6. \* Describe any potential for direct social impact in this study . For example, any engagement with specific the specific communities if applicable:

decrease the mortality rate due to cervical cancer, however, these valuable tools are not used in adequate rates by the Evidence shows that cervical cancer prevention methods such as screening and getting HPV vaccine are essential to Muslim community. Therefore, understanding the Muslim women's behaviors and offering an educational program to provide individuals with crucial insight into these tools.

## 7. Upload a supporting citation list if applicable:

| | Document<br>Name | Document | Version | Version Date Upl<br>Modified By | Uploaded <sub>Type</sub><br>I By | Туре | Approved |
|---|---|---|---|---|---|---|---|
| View | View Consent form focus group | Namoos- Consent 0.03<br>from of focus<br>group<br>05.12.2023.pdf | 0.03 | 7/8/2023<br>1:09 AM | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | Yes |
| View | Consent form -<br>Intervention<br>program | View Consent form - Namoos- Consent 0.04 Intervention from of Intervention group 05.12.2023 copy.pdf | 0.04 | 7/8/2023<br>1:09 AM | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | Yes |
| View | View Fund Plan | Asmaa -Budget<br>04.13.2023.xlsx | 0.03 | 5/12/2023 Asmaa<br>11:52 AM Namoo | Asmaa<br>Namoos | Funding Proposal | Not<br>Applicable |
| View | View Education<br>session | Asmaa Education 0.02 session guide, intervention group-04.07.2023.docx | 0.02 | 5/12/2023 Asmaa<br>10:52 AM Namoos | Asmaa<br>Namoos | Other | Yes |

| t Version Date Modified eline 0.02 5/12/2023 | Version Date Modified 0.02 5/12/2023 | sion Date<br>Modified<br>5/12/2023 | Date Uploader<br>Modified By<br>5/12/2023 Asmaa | Uploade<br>By<br>Asmaa | 70 | <b>Type</b><br>Other | Approved |
|---|---|---|---|---|---|---|---|
| for PROMIS 10:43 AM women Projectdocx | s, uneille 0.02 3/12/2023 DMIS 10:43 AMdocx | 10:43 AM | | Namoos | | | 80 |
| Conceptual Asmaa 0.02 5/12/2023 Asmaa model Conceptual Model 10:40 AM Namoos 05.12.2023.docx | 0.02 5/12/2023<br>el 10:40 AM | 5/12/2023<br>10:40 AM | | Asmaa<br>Namoos | | Research Measure | Yes |
| Flayer 2 Asmaa Flyer 0.01 5/12/2023 Asmaa<br>Version 10:39 AM Namoos<br>05.12.2023.docx | Flyer 0.01 5/12/2023 10:39 AM 10:39 AM 123.docx | 5/12/2023<br>10:39 AM | , | Asmaa<br>Namoos | | Other | Yes |
| Namoos-Focus Namoos -Focus 0.02 5/12/2023 Asmaa group script Group Script 10:24 AM Namoos guide Guide.docx | Namoos -Focus 0.02 5/12/2023<br>Group Script 10:24 AM<br>Guide.docx | 5/12/2023<br>10:24 AM | 1 | Asmaa<br>Namoos | | Other | Yes |
| Participants -RA Namoos- 0.01 5/12/2023 Asmaa communication Participants -RA 6:45 AM Namoos script communication script docx | 0.01 5/12/2023 , and a second of the second | 5/12/2023<br>6:45 AM | ო<br>ი | Asmaa<br>Namoos | vo. | Other | Yes |
| Study Survey( Survey- Promise 0.01 5/12/2023 Asmaa Pre-post and women project 6:35 AM Namoos satisfactory 05.12.2023.docx scales) | 0.01 5/12/2023 6:35 AM | 5/12/2023<br>6:35 AM | , | Asmaa<br>Namoo | Ø | Research Measure | Yes |
| consent form- Consent from - 0.01 2/20/2023 Asmaa focus group 4:32 PM Namoos 02.20.2023.docx | 0.01 2/20/2023 ,<br>4:32 PM | 2/20/2023 .<br>4:32 PM | ` - | Asmaa<br>Namoo | v | Consent/Assent/Information No<br>Sheet | oN r |
| View VS biosketch Sheppard 0.01 2/20/2023 Asmaa Biosketch for AN 4:00 PM Namoos 11.14.2022.pdf | 0.01 2/20/2023 ,<br>for AN 4:00 PM<br>2.pdf | 2/20/2023 ,<br>4:00 PM | <b>,</b> – | Asmaa<br>Namoos | " | CV/Biosketch | Not<br>Applicable |
| Communication Communication 0.01 2/20/2023 Asmaa log log.docx 3:59 PM Namoos | Communication 0.01 2/20/2023 log.docx 3:59 PM | 2/20/2023<br>3:59 PM | | Asmaa<br>Namoos | | Other | Yes |
| PRMC approval 2022-10- 0.01 10/10/2022 Asmaa 10_MCC-22- 12:30 PM Namoos 19873_PRMC Approval Letter.pdf | 2022-10- 0.01 10/10/2022<br>10_MCG-22- 12:30 PM<br>19873_PRMC<br>Approval<br>Letter.pdf | 10/10/2022<br>12:30 PM | | | (0 | Ancillary Committee<br>Approval | Not<br>Applicable |
| Flyer 0.01 4/8/2022 Asmaa 004.08.2022.png 6:09 PM Namoos | 0.01 4/8/2022<br>8.2022.png 6:09 PM | 4/8/2022<br>6:09 PM | - | Asmaa<br>Namoo | Ø | Other | Yes |
| Namoos Dr. Namoos A. 0.01 4/3/2022 Asmaa<br>Resume Biosketch 3:47 PM Namoos | 0.01 4/3/2022 ,<br>3:47 PM | 4/3/2022<br>3:47 PM | , _ | Asmaa<br>Namoo | Š | CV/Biosketch | Not<br>Applicable |

HM20024502

7/8/23, 9:07 AM

Document Document V

Version Date Uploaded Type Modified By

Approved

View: SF2 - Study Population HM20024502 ID: HM20024502

## PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

## Study Population

- 1. \* Provide the maximum number of individuals that
- 1. May participate in any study interaction or intervention (Including screening, consenting, and study activities

AND/OR

2. You obtain any data/specimens about (regardless of identifiability)

at VCU and at other sites under the VCU IRB's oversight. See the help text for additional guidance.

- 2. If this is a multi-Center Project, what is the maximum anticipated number of subjects across all sites?
- participants. The team members will approach potential respondents at Islamic centers to participate in this study. The nclusion criteria include women aged ≥18 years who speak English, self-identify as Muslim, and have not participated in our pilot study before. The exclusion criteria are any participants who participated in our pilot study or are unable to Sample: A non-probability sampling (convenience sampling) method will be adopted to allow reach all potential 3.  $^{st}$  Provide justification for the sample size by explaining how you arrived at the expected number of participants and why this number is adequate for answering the research questions provide valid consent (e.g., developmental disability).

Qualitative analysis side: to develop the education material we will recruit 10 female participants above 18 years old content to achieve each target (design). As a next step the focus group will focus on the formatting of the material including basic usability testing (refine). Based on information from these sessions we will finalize the educational materials for the intervention. First the focus group will help select the targets of the proposed education and the who identify as Muslim to participate in the design of the religiously tailored and culturally appropriate education material for our intervention.

we will use the grounded theory for complete the analysis

software sample size calculator for the minimal sample size needed for an unlimited population size using a confidence 10% post-intervention. Based on a power analysis assuming the use of the student T-test to assess the difference in Statistical Analysis for quantitative side: We assume that our study's CC-S HPV-Vax uptake rate would increase by outcome between the intervention and control groups, The target sample size is estimated based on the G power interval of 80%, a standard deviation of 0.5, and a margin of error of 5%. The study requires 10 participants for intervention to test the feasibility of the program.

ntervals will be reported to convey the precision of all point estimates. Following the descriptive analyses, comparisons attitudes, and risk perceptions of CC-S and attitudes and intention to get the HPV-Vax. Means, standard deviations, Summaries will be stratified by gender, age, education, language, and community to explore patterns. Confidence Descriptive summaries will be generated to summarize participant demographics and all study variables including and percentiles will be reported for continuous variables, frequencies, and percentages for categorical variables. individual and community characteristics, with a particular focus on religious adherence, modesty, knowledge,

defined by gender, age, religion, education, language, and community. We will use ANOVAs and t-tests for continuous multiple linear regression analysis after log transformation of the knowledge score. A statistically significant difference will be made to identify differences in knowledge, attitudes and risk perceptions, and HPV-Vax intent between groups Bonferroni) will follow significant omnibus ANOVA results to determine which groups differ while controlling the Type-I assumptions of parametric methods. The relationship between the knowledge score and the independent categorical variables (e.g., perceived risk and attitudes) and Chi-square tests for categorical variables). Post-hoc tests (Tukey's, error rate. Non-parametric alternatives (e.g., Fisher's exact test, Kruskal-Wallis) will be used if data do not meet the multinomial variables. Variables that were significantly associated with the knowledge score were included in the variables was determined using the Mann–Whitney U test for binomial variables and the Kruskal–Wallis test for will be defined as a p-value was less than 0.05. Data analysis will be conducted using the R program.

## 4. \* List the study inclusion criteria:

-For focus group to test the education material ( n= 10 focus group)

The inclusion criteria include women aged ≥18 years who speak English, self-identify as Muslim, are able to give valid consent, who not participated in our pilot before.

-For Intervention program (n=20)

The inclusion criteria include women aged ≥18 years who speak English, self-identify as Muslim, are able to give valid consent, who not participated in our pilot and focus group before

We will use 4 centers at the time of recruitment: the Islamic center of Richmond, the Islamic center of Henrico, the Islamic center of Hampton, and the Peninsula Islamic Community Center

## 5. \* List the study exclusion criteria:

Phase 1)

Aim 1 a and b

-ormative research-focus group

Sample size: 10 Muslim women

Sampling: Purposeful sampling.

Inclusion criteria:

-Female Muslim individuals above 18 years old.

-Able to speak and understand English

-Have not had a hysterectomy.

Have not had a cervical cancer diagnosis.

-Willing to participate in the educational program and undergo cervical cancer screening.

Physically well, able to give consent form

Phase 2

Aim 2 and 3

Single arm trial - pre and post-test

Sample size: 20 Muslim Women.

Sampling: Non-probability sampling (convenience sampling)

nclusion criteria:

Female Muslim individuals above 18 years old.

-Able to speak and understand English. Have not had a hysterectomy.

-Have not had a cervical cancer diagnosis

 Willing to participate in the educational program. Physically well, able to give consent form

·Have not participated in our pilot study before

We will be excluded any participant who was recruited during our pilot study (IRB: HM20021579).

7. Justify the inclusion and exclusion criteria if you are either targeting, or excluding, a particular segment of the population / community. Provide a description of the group/organization/community and provide a rationale.

We are excluding non-English speakers because: 1 There is insufficient budget to hire other language speakers.

2. The Muslim population is very diverse, and it isn't easy to include all languages. 3. Translating the study material and aims will affect the study quality.

HM20024502 ID: HM20024502 View: SF2 - Background, Rationale & Goals Section Complete

PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn HM20024502 - Vanessa Lavene Sheppard methods among Muslim Americans WOMEN

# Background, Rationale & Goals Section Complete

Protocol Progress:

- **INITIAL SETUP**
- **■** BACKGROUND, RATIONALE & GOALS

- (a) RESEARCH PLAN (b) CONSENT PLAN (c) RISKS, PRIVACY & CONFIDENTIALITY (c) POPULATIONS WITH SPECIAL CONSIDERATIONS (7) INSTITUTIONAL REQUIREMENTS (8) DOCUMENTS

Click Continue below to go to the next section

ID: HM20024502

HM20024502 View: SF2 - Study Procedures

## PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

## Study Procedures

Aim 1b. We will conduct individual interviews with key stakeholders in our Community Advisory Board (Muslim religious leaders (N=4)) to receive feedback on the developed materials and inform the intervention program. This aim includes 1. \* Describe the study hypothesis and/or research questions. Use lay language whenever possible. he Phase II (Preliminary Testing) of the ORBIT model (proof of concept, prepare the pilot)

acceptance of cervical cancer screening and prevention. This aim includes the Phase III (Efficacy) of the ORBIT model participants with the same eligibility criteria as in Aim 1, who have not participated in our previous studies, and conduct a single-arm pilot trial. H2. We hypothesize that the religiously tailored and culturally appropriate intervention program H1. Participants will show significant improvements in knowledge and acceptance of cervical cancer prevention after Aim 2. We will test the preliminary efficacy of the religiously tailored and culturally appropriate intervention program. will be feasible to conduct as evidenced by meeting enrollment targets and the ability to implement the program as planned. H3. The intervention will be acceptable as evidenced by engagement (>60%) and retention (>80%), and the intervention. To test this hypothesis, we will conduct a pre-post survey to examine changes in knowledge and Aim 3. We will test the feasibility and acceptability of the religiously tailored and culturally appropriate intervention program which includes education and experiential practice/communication skills training. We will recruit 20 satisfaction survey ratings.

2. \* Describe the study's specific aims or goals. Use lay language whenever possible.

competency of healthcare providers related to the Muslim culture at the VCU health system. Our ongoing work with the methods. The secondary outcome is the acceptability and confidence/trust in cervical cancer prevention methods such and HPV-Vax. The Muslim Community Partners (MCPs) will collaborate with our institute (VCU) by reaching out to four Muslim community has informed us about the community's needs. In this project, we will implement an interventional motivator for Muslim families to change. The primary outcome is increasing awareness of cervical cancer prevention interventions, which combine health-related religious teachings and scientific information about the benefits of CC-S convince women to join our study, reach out to a high number of MAW, and because religious voices will be a good Islamic religious centers in Virginia. Partnership with Islamic centers is valuable to our project due to their: ability to program guided by a community-based participatory approach utilizing expert-led education sessions and peer-led Our team also investigates the barriers faced by MAW in the US healthcare system by evaluating the cultural

The research questions are: Would MAW intend to do cervical cancer screening and uptake the HPV Vaccination after an education program supported by the Mosques that they frequently visit?

The aims of the study are:

Aim 1b. We will conduct individual interviews with key stakeholders in our Community Advisory Board (Muslim religious leaders (N=4)) to receive feedback on the developed materials and inform the intervention program. This aim includes Aim 2. We will test the preliminary efficacy of the religiously tailored and culturally appropriate intervention program. he Phase II (Preliminary Testing) of the ORBIT model (proof of concept, prepare the pilot).

 $https://irb.research.vcu.edu/irb/app/portal/smartform/printProject/\_Protocol/7B0E834A95711ECC991CBE9AD565000?packetIds=defaultPrintPacket$ 

acceptance of cervical cancer screening and prevention. This aim includes the Phase III (Efficacy) of the ORBIT model participants with the same eligibility criteria as in Aim 1, who have not participated in our previous studies, and conduct a single-arm pilot trial. H2. We hypothesize that the religiously tailored and culturally appropriate intervention program H1. Participants will show significant improvements in knowledge and acceptance of cervical cancer prevention after will be feasible to conduct as evidenced by meeting enrollment targets and the ability to implement the program as planned. H3. The intervention will be acceptable as evidenced by engagement (>60%) and retention (>80%), and Aim 3. We will test the feasibility and acceptability of the religiously tailored and culturally appropriate intervention he intervention. To test this hypothesis, we will conduct a pre-post survey to examine changes in knowledge and program which includes education and experiential practice/communication skills training. We will recruit 20 satisfaction survey ratings.

For these aims, we will use a survey that includes:

Pre-test survey, the scales are:

- Demographic
- 2. Perceived Discrimination
  - 3. Religious Discrimination
- Spiritual Health Locus of Control.
  - 5. Modesty
- 6. Cervical Cancer Knowledge
  - 7. Perceived risk
    - 8. Cuse of action
      - 9. Self-efficacy
- 10. Attitude about CC screening
- 11. HPV vaccination acceptability

Prost-test survey, the scales are:

- 2. Perceived Discrimination
- 3. Religious Discrimination
- Spiritual Health Locus of Control.
  - 5. Modesty
- Gervical Cancer Knowledge
- Perceived risk
- 8. Cuse of action
- Attitude about CC screening
- 10. HPV vaccination acceptability
- 11 General Self-Efficacy Scale (GSES)
- 12. Cervical Cancer Screening Self-Efficacy Scale

Satisfactory survey are:

- -Experience with the intervention.
- Acceptability of content
- -Acceptability of delivery

| | E-mail invitations |
|---|----------------------------------------------------------------------|
| | Phone Solicitation scripts (i.e. cold calls or random-digit-dialing) |
| > | Flyers, Mailed Letters or Newspaper/TV/Radio Ads |
| | TelegRAM announcements |
| | Website text |
| | Study-specific web sites (provide the design and text) |
| | Social Media |
| | EPIC MyChart Patient Portal research study descriptions |
| | Psychology Research Participant Pool (SONA) study descriptions |
| | Scripts for announcements made to groups |
| | Other recruitment document |
| | No recruitment materials |

- 4. \* Describe the study procedures/methods for identifying and recruiting participants. Address all of the following three aspects of recruitment in your response.
- Identification of potentially eligible participants or secondary data/specimens of interest. - What database(s) will be queried to identify secondary data/specimens
- How VCU Informatics or VCU IRDS will be used for cohort identification (when applicable, see help text)
  - How potential participants' contact information will be obtained
- 2. Recruitment procedures to invite participation in the study (when applicable):
- How each of the written or verbal recruitment materials and reminders (selected above) will be used
  - Who will contact, approach, or respond to potential participants - Locations where recruitment procedures will take place
    - The timing and frequency of recruitment attempts
- 3. Eligibility screening prior to consent and how those activities will be carried out (when applicable)

## See the help text for additional guidance.

The principal investigator (PI) has a community partnership with the Islamic Center of Richmond, where the research predetermined times where women could approach study team members to ask questions, sign up for participation, team will distribute flyers about the project (see attachment). The research team will be present at the Mosque at and schedule appointments.

- 1) Identification of potentially eligible participants:
- -The research team will distribute flyers about the project at the Islamic Center of Richmond to identify potentially eligible participants.
- -The education material will be mentioned as PDF in the docs section
- 2) Recruitment procedures to invite participation in the study:

Participants: Women interested in participating can approach study team members to ask questions, sign up for Place: The research team will be present at the Mosque during predetermined times. participation, and schedule appointments.

The research assistant will handle contact with potential participants, including scheduling interviews and baseline verbal recruitment materials will be used when study team members interact with potential participants. Written recruitment materials, such as flyers, will be distributed to provide information about the study.

Recruitment procedures will take place at the Islamic Center of Richmond.

3) Eligibility screening prior to consent and how those activities will be carried out:

For the one-arm clinical trial, participants will be screened for eligibility during the scheduling of baseline surveys. During these interactions, eligibility screening will be conducted to ensure participants meet the study criteria. For focus group meetings, participants will be screened for eligibility before being scheduled for interviews. The research team will use a standardized screening tool or questionnaire to assess eligibility

The survey will be given to the potential participants in person ( hard) or through QR code through redcap

The education materials will be clearly outlined in the study plan PDF.

Summary the intervention:

sections/videos. The session will be offered in a single day and last 1.5 hours. The session will include the following topics: 1) Risk of HPV infection (30 minutes), 2) Cervical cancer risk (30 minutes), and 3) Advantages and benefits of The intervention group will consist of 20 participants who will receive one education session divided into three early screening and the HPV vaccine (30 minutes)

material. The survey will be self-report, available in both hard copy and electronic form with a QR code for Redcap. All participants from both groups will be given the survey at month 0 (baseline) after the delivery of the educational

Participants are expected to take approximately 45 minutes to complete the survey.

The Islamic center offer private room to practice the research activities in both phases ( Focus group and single arm

5. \* Does this study have a separate protocol document (i.e. a multisite or sponsor's protocol) that contains a detailed description of the study's methodology?



)

understandable to those IRB committee members whose expertise is not scientific. The description must 6. \* Since a separate protocol document is not uploaded, describe the proposed research using language

- 1. A statement explaining the study design
- 2. A detailed description of all the procedures that will be followed to carry out the study, preferably in sequential order, and in sufficient detail that the study's methods could be replicated
- 3. The schedule and frequency of when and how procedures will be conducted (e.g. in person, online, phone,
- 4. A description of all research measures/tests/interventions that will be used, including analyses/tests conducted on specimens/biological samples (if applicable)

## See the help text for additional guidance

A statement explaining the study design

Study Design:

The proposed study consists of two parts.

Part 1 involves formative research through a focus group to gather insights and reach saturation. Part 2 is a single-arm pre and post-test trial with the objective of evaluating the efficacy of an educational interventional

The study aims to increase cervical cancer screening (CC-S) and HPV vaccine (HPV-Vax) rates among Muslim American women (MAW) in Virginia, leading to a reduction in cervical cancer (CC) incidence and mortality

- A detailed description of all the procedures that will be followed to carry out the study, preferably in sequential order, and in sufficient detail that the study's methods could be replicated.
- a. Part 1 Formative Research: Conduct a focus group with 10 participants until saturation is reached.
- b. Part 2 Single-arm Pre and Post-test Trial: Enroll 20 participants to evaluate the educational program's effectiveness

Participants will complete a baseline survey to assess their knowledge, attitudes, CC-S and HPV-Vax practices, and predisposing factors.

The survey will cover topics such as CC knowledge, experiences of medical mistrust, discrimination, spiritual coping,

3. The schedule and frequency of when and how procedures will be conducted (e.g. in person, online, phone, paper,

All procedures will be conducted in person at the Islamic Centers, except for follow-up phone calls.

Recruitment will occur during regular Friday prayers and religious holidays.

Participants will receive a brochure explaining the study and be screened for eligibility by the Research Assistant (RA). Eligible participants will be given a telephone contact for enrollment at a more convenient time.

The consent process will involve verbal explanation, providing the consent form in English, and allowing participants to

Follow-up surveys and confirmations will be conducted via phone calls.

4. A description of all research measures/tests/interventions that will be used, including analyses/tests conducted on specimens/biological samples (if applicable) Power Analysis: No power analysis for this study, A target sample size of 20 participants has been determined based on PhD committee, the purpose of the project is training for the STUDENT

Measures: Validated scales and surveys will be used to measure

Age: Age can be measured using a simple demographic question such as "What is your age?" in the pre- and postintervention surveys. Education: Education level can be measured using a simple demographic question such as "VVhat is the highest level of education you have completed?" in the pre- and post-intervention surveys.

Modesty and Conservatism: can be measured using a combination of demographic questions and attitudinal scales. conservative would you describe yourself?" while attitudinal scales could include items such as "I am comfortable discussing reproductive health issues with my healthcare provider" or "I am willing to discuss cervical cancer ☐ For example, demographic questions could include "How important is modesty in your culture?" or "How prevention activities with my family and friends."

you ever had a Pap smear?" or "Have you ever received the HPV vaccine?" in the pre- and post-intervention surveys. Cervical Cancer Screening and HPV Vaccine Uptake: can be measured using self-reported questions such as "Have Additional questions can also be included to determine the frequency and timing of screening and vaccine uptake.

Participants' Knowledge and Attitude: can be measured using a combination of open-ended and closed-ended

ended questions could include "Do you believe that cervical cancer screening is important?" or "Do you believe that the □Open-ended questions could include "What do you know about cervical cancer prevention activities?" while closed-HPV vaccine is safe and effective? Feasibility of Intervention: can be measured by tracking enrollment rates, attendance rates, and completion rates in the pre- and post-intervention surveys.

Additional questions can also be included to assess the overall acceptability of the intervention among participants.

Self-efficacy: can be measured using a self-efficacy scale specific to cervical cancer screening, such as the Cervical Cancer Screening Self-Efficacy Scale (CCSES), as described in the previous answer

survey could include questions such as "Did you find the program useful?" or "Would you recommend this program to a Acceptability of the Program: can be measured using a satisfaction survey at the end of the intervention program. The

#### Outcomes

Secondary outcomes include an increase in knowledge and awareness, an increase in self-efficacy, and improvement The primary outcome in increase the number of women who undergo cervical cancer screening. in attitudes towards cervical cancer prevention.

Long-term outcomes include a reduction in cervical cancer incidence and mortality, sustainability of behavior change, and a reduction in healthcare costs associated with advanced-stage cancer treatment.

Moderator factors that can influence the effectiveness of the program include age, education level, ethnicity, socioeconomic status,

Mediating mechanisms that explain how the program leads to its outcomes include improved knowledge and awareness, increased self-efficacy, attitude change, increased and social support, Identifying and addressing moderator factors and mediating mechanisms can help to tailor the program to the specific needs and preferences of the target population and maximize its effectiveness

7/8/23, 9:07 AM

HM20024502

Key Study Variables: Socio-demographic variables, cultural/religious practices, cancer literacy, knowledge, perceived isk, barriers, benefits, and participation in preventive measures.

Evaluation Measures: Intervention acceptance will be self-reported, covering challenges, barriers, facilitators, likes/dislikes, and suggestions for improvement.

involving in-person procedures, phone follow-ups, and self-report measures. The proposed methods are designed to evaluate the effectiveness of the educational program and its impact on CC-S and HPV-Vax rates in the target sequential approach of formative research and a single-arm trial. The study will be conducted at Islamic Centers, This study aims to address barriers to CC prevention among MAW through an educational intervention, using a

These tests will help determine whether there are statistically significant differences between the pre- and post-survey Statistical Tests: Statistical tests such as t-tests or ANOVA can be used to analyze the data from the pre-post survey. results and whether the intervention had a significant effect on participants' knowledge and acceptance of cervical cancer prevention.

- 7. \* The IRB only reviews research activities, so indicate for each of the study activities described in the question above or in the protocol which activities are:
- Being performed exclusively for research purposes (i.e. they would not otherwise be done apart from this study) VERSUS.
- Alterations of routine activities/procedures (e.g. the study is altering the timing, frequency, method location, amount, etc.) VERSUS.
- Being done for other purposes and whose data/results will be used secondarily in the study (e.g. standard medical or psychological tests, routine education practices, quality improvement initiatives, etc.) See the help text for additional guidance

The study is being performed exclusively for research purposes.

- 8. If applicable, describe alternatives (research or non-research) that are available to potential participants if they choose not to participate in this study:
- 9. Upload any supporting tables or documents (e.g. protocol documents, figures/tables, data collection forms, study communications/reminders)

Upload ALL instruments/guides that will be used or that participants will experience (i.e. see, hear, complete), including measures, scripts/questions to guide interviews, surveys, questionnaires, observational guides, Upload ALL recruitment and screening materials, including such as ads, flyers, telephone or in-person scripts, letters, email invitations, TelegRAM announcements, and postcard reminders, screening scripts, screening forms, and screening measures:

| t Version Date Uploaded Type Approved<br>Modified By | nsent 0.03 7/8/2023 Asmaa Consent/Assent/Information Yes<br>1:09 AM Namoos Sheet |
|---|---|
| Document | Namoos- Consent 0.03 7/8/2 from of focus 1:09 |
| Document<br>Name | View Consent form focus group |

HM20024502

7/8/23, 9:07 AM

| | Document<br>Name | Document | Version | Date<br>Modified | Version Date Uploaded Type Modified By | Туре | Approved |
|---|---|---|---|---|---|---|---|
| View | View VS biosketch | Sheppard<br>Biosketch for AN<br>11.14.2022.pdf | 0.01 | 2/20/2023 Asmaa<br>4:00 PM Namoos | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |
| View | View Communication Communication log log-docx | Communication log.docx | 0.01 | 2/20/2023 Asmaa<br>3:59 PM Namoos | Asmaa<br>Namoos | Other | Yes |
| View | View PRMC approval 2022-10-10-10-10-10-10-10-10-10-10-10-10-10- | 2022-10-<br>10_MCC-22-<br>19873_PRMC<br>Approval<br>Letter.pdf | 0.01 | 10/10/2022 Asmaa<br>12:30 PM Namoos | Asmaa<br>Namoos | Ancillary Committee<br>Approval | Not<br>Applicable |
| View | View F <b>lyer</b> | Flyer<br>004.08.2022.png | 0.01 | 4/8/2022<br>6:09 PM | Asmaa<br>Namoos | Other | Yes |
| View | View Namoos<br>Resume | Dr. Namoos A.<br>Biosketch<br>06.07.2021.pdf | 0.01 | 4/3/2022<br>3:47 PM | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |

View: SF2 - Project Details HM20024502 ID: HM20024502

## methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn

### **Project Details**

An intervention includes both physical procedures by which information or biospecimens are gathered (e.g., venipuncture) and manipulations of the subject or the subject's environment that are performed for research purposes.

An interaction includes communication or interpersonal contact between investigator and subject. It may include in-person, online, written, or verbal communications.

Secondary information/biospecimens are information or biospecimens that have been or will be collected for some other "primary" or "initial" activity and that will be used secondarily in the research study.

| 1. * Sele | * Select all of the following types of interventions that apply to this study (selections will branch): |
|---|---|
| > | Social/Behavioral interventions or experimentation / Tasks / Environmental manipulations |
| | Deception (misleading participants through false or incomplete information) |
| | Drug(s) / Biologics / Supplement(s) / Other Compounds (investigational products or products whose administration is dictated by the study protocol and not per the physician's clinical judgment) |
| | IV contrast administration for research-related imaging (will branch to the Drugs page) |
| | Placebos |
| | Safety and/or effectiveness evaluation of Bio-Medical Device(s), including in-vitro diagnostic devices/assays, mobile medical apps, software functions, and HUDs used in clinical investigations |
| | Washout Periods |
| | Expanded Access – Treatment Use of an Investigational Product |
| | Medical or Surgical Procedures (eg: physical exam, clinical procedures, scans, etc) |
| | Specimen/biological sample collection |
| | None of the Above |

Active Internet data collection (i.e. using the internet to collect data, including online surveys, data 2. \* Select all of the following types of interactions and methods of data collection that apply to this study Surveys / Questionnaires /Written responses to questions (including data entry) Passive Internet data collection (i.e. passively observing online behavior, bots) Interviews / Focus Groups / Verbal responses to questions Audio / Video recording or photographing participants Educational Settings/Assessments/Procedures 3. \* Select all types of recordings that will be made: collection via Zoom, apps, etc.) None of the Above (selections will branch): Observations Audio Video

4. \* Describe the purpose of the recordings, who will be recorded and when such recordings will occur:

**Photographs** 

be used to transcribe the data and analyze the transcripts. The research assistant conducting the interviews will record The recordings in Part 1, which involve the focus group interviews, are for analysis purposes. The audio recordings will important to note that the research assistant will not use any names or identification during the interviews to ensure the sessions using a VCU iPad. The interviews will take place in the private room provided by the mosque. It's confidentiality

Part 2:

community outreach work. These photos will be used exclusively for conference purposes to disseminate the findings In Part 2, the recordings serve a different purpose. During the education sessions, photos will be taken as part of the of the study. Similar to Part 1, the research assistant will use a VCU iPad to record the sessions, but no identifying information will be used or captured during the interviews.

using a VCU iPad in the private room provided by the mosque, and precautions are taken to ensure confidentiality and the recordings are used to facilitate analysis in Part 1 and for dissemination purposes in Part 2. They are conducted anonymity of the participants.

5. \* Select all types of secondary information and/or specimens that apply to this study (selections will branch) See the help text for definitions.  $https://irb.research.vcu.edu/irb/app/portal/smartform/printProject/_Protocol/7B0E8344A95711ECC991CBE9AD565000?packetIds=defaultPrintPacket$ 

7/8/23, 9:07 AM

HM20024502

ID: HM20024502

View: SF2 - Behavioral Intervention/Task Details

## HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN

## Behavioral Intervention/Task Details

This page asks for details about the social/behavioral intervention, task, or environmental manipulation in the research.

Interventions include both physical procedures by which information is gathered and manipulations of the subject or the subject's environment that are performed for research purposes. This might include activities such as playing computer games, performing a task, thought/cognition activities, environmental manipulations, and educational activities. If the study only involves surveys, interviews, or secondary data collection, go back to the Project Details page and uncheck 'Social/Behavioral interventions or experimentation / Tasks / Environmental manipulations" in Question 1.

- 1. \* Describe the duration of the social/behavioral intervention, task, or environmental manipulation: The event will be organized for three hours
  - The education sessions will be 1.5 hours (90 minutes).
  - I ne education sessions will be 1.5 nours ( 90 mir - The self-report survey will take 45 minutes.
- The rest of the time, we will have a break and lunch.

The education sessions will be offered on Saturday and Sunday.

- 2. \* Describe any potential harms or discomforts that participants could experience during the intervention activity:
- They may experience some psychological discomfort related to some of the questions. Participation in research might nvolve some loss of privacy. There is a small risk that someone outside the research study could see and misuse nformation about you.
- 3. \* Will the intervention activity be physically invasive or painful?



S N

- 4. \* Describe the impact the intervention activity will have on participants, including the nature and duration of any impact(s):
  - There is no impact on the intervention process except for the cultural sensitivity that we mentioned before.
- 5. \* In the investigator's opinion, is there any reason to think that the participants will find the intervention activity offensive or embarrassing? Explain why or why not.
  we have been working with this community for three years, and we don't feel that there is any offensive or
View: SF2 - Active Internet Data Collection HM20024502 ID: HM20024502

### PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

## Active Internet Data Collection

internet. If proposing a non-VCU approved platform, give the rationale for selecting the technology instead of 1. \* Describe the platform/technology chosen for collecting the data and transmitting data securely over the a VCU-approved platform.

is a widely used, secure, and HIPAA-compliant web-based application specifically designed for research data collection The chosen platform for collecting survey data in this study is REDCap (Research Electronic Data Capture). REDCap and management. It provides a user-friendly interface for designing surveys, capturing data, and generating reports.

devices offer built-in voice recording features that can be used by the research assistant during interviews or other data For note recording, the Apple system will be utilized, likely referring to Apple devices such as iPads or iPhones. These collection activities.

reliable tool for research data. It is designed to meet rigorous data protection standards, ensuring the privacy and confidentiality of participants' information. Additionally, REDCap offers a range of features for data validation, quality The rationale for selecting REDCap as the survey collection platform is its established reputation as a secure and control, and export options, which contribute to efficient and accurate data management.

policies, the decision to utilize REDCap and the Apple system may stem from specific functionalities and familiarity with these technologies. Researchers may have found that these platforms meet their data collection and recording needs While using a VCU-approved platform is typically encouraged to maintain consistency and alignment with institutional effectively, and they have confidence in their security and reliability.

# 2. \* Describe how data will be linked or unlinked to identifiers including email addresses, names, and/or IP

that personal identifying information, such as names and email addresses, will not be linked to their survey responses. Instead, each participant will be assigned a unique study ID or code, which will be used to anonymize their data. This For the survey data collected through the REDCap platform, participants' responses will be de-identified. This means any names or identification during the interviews. This further ensures that participants' personal information remains Regarding the note recordings using the Apple system, it is important to note that the research assistant will not use In this study, data will be collected and stored in a manner that ensures the protection of participants' confidentiality and privacy. Specifically, data will be unlinked from identifiers such as email addresses, names, and IP addresses. separation of identifiers from survey responses helps maintain the confidentiality of participants' information. unlinked from the recorded data.

By unlinking data from identifiers, the study aims to protect participants' privacy and confidentiality throughout the data collection and analysis process. It reduces the risk of unauthorized access or disclosure of sensitive information, promoting ethical research practices.

## How will you protect your data collection from fraudulent responses:

- 1. Collection of IP addresses: we are not collecting IP address
- 2. Identity verification procedures: Implementing procedures to verify participants' identities can add an extra layer of

protection against fraudulent responses. This can include requesting additional identification information or using verification methods like email confirmation.

- meet the eligibility criteria or who provide inconsistent or implausible responses. These questions can help ensure that Screening questions: Including screening questions within the survey can help filter out respondents who may not only qualified and genuine participants are included in the study
  - 4. Attention checks: Incorporating attention check questions within the survey helps assess the attentiveness and sincerity of participants. These questions are designed to identify respondents who may be providing random or careless responses. Participants who fail attention checks may be excluded from the analysis.
- 5. Post-data collection monitoring procedures: Regularly reviewing and monitoring the collected data can help identify any suspicious or fraudulent responses. Data quality checks, including identifying outliers or patterns of unusual responses, can be conducted to ensure the integrity of the data

collected. It is essential to consider the specific needs of the study and balance the level of protection with the potential combination of these strategies can help safeguard against fraudulent responses and protect the validity of the data While the specific protections employed will depend on the nature and requirements of the study, implementing a mpact on participant engagement and response rates.

## 4. $^{*}$ Is there an alternative method for completion of the data collection other than the internet?



ŝ

5. \* Describe how individuals will be able to skip or not answer particular questions. If any questions are mandatory, provide justification.

nstrument will be designed in a way that allows participants to proceed through the questionnaire without being In the study, participants will be provided with the option to skip or not answer particular questions. The survey equired to answer every single question. The following approach will be implemented:

- choose whether or not to answer them. This allows participants to skip questions that they may feel uncomfortable with 1. Optional Questions: The majority of questions in the survey will be designed as optional, meaning participants can or prefer not to answer. They can simply move on to the next question or section of the survey
  - 2. Mandatory Questions: In some cases, certain questions may be designated as mandatory. These questions will be mandatory questions will be provided in the study design and protocol documentation, explaining the importance of carefully selected based on their criticality to the research objectives or eligibility criteria. Justification for including obtaining specific information for the study outcomes or participant eligibility.
- 3. Justification for Mandatory Questions: The justification for including mandatory questions will be based on scientific intervention's effectiveness. Additionally, if certain eligibility criteria need to be met for participant inclusion, mandatory or practical reasons. For example, if the study aims to assess the impact of a specific intervention on a particular variable, it may be necessary to include mandatory questions related to that variable to accurately evaluate the questions may be necessary to determine if individuals meet those criteria.
  - Allowing participants to skip or not answer particular questions, the study respects participant autonomy and ensures hat their comfort and privacy are prioritized. Mandatory questions are justified based on research objectives or eligibility criteria, ensuring that the necessary information is collected to achieve the study's goals.

# If not including children, describe any procedures used to verify that research participants are adults.

providing valid identification documents, such as a driver's license or passport, which clearly indicate their date of birth. To ensure that research participants are adults and meet the eligibility criteria, specific procedures will be implemented verification process will help ensure the accuracy and integrity of the study data, as well as maintain compliance with to verify their age. During the recruitment process, potential participants will be required to confirm their age by The research team will review and verify these documents to confirm that participants are indeed adults. This ethical considerations related to involving adult participants in the research.

HM20024502

ID: HM20024502

View: SF2 - Costs to Participants

### methods among Muslim Americans WOMEN PROMIS WOMAN Education Program: ImProving ceRvical cancer prevention HM20024502 - Vanessa Lavene Sheppard

### Costs to Participants

| 1. * Sele | 1. * Select all categories of costs that participants or their insurance companies will be responsible for: |
|---|---|
| > | Participants will have no costs associated with this study |
| | Study related procedures that would be done under standard of care |
| | Study related procedures not associated with standard of care |
| | Administration of drugs / devices |
| | Study drugs or devices |
| | Other |

View: SF2 - Compensation HM20024502 ID: HM20024502

### methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn

### Compensation

(monetary or non-monetary) to the IRB to ensure the plan will comply with VCU policies. Refer to WPP XVII-2 for the IRB's It is recommended that investigators consult with VCU Procurement Services before proposing a compensation plan guidelines about compensating research participants.

- Describe any compensation that will be provided including:
  - 1. total monetary amount
- type (e.g., gift card, research pre-paid card, cash, check, merchandise, drawing, extra class credit)how it will be disbursed
- 4. how you arrived at this amount
- 5. What identifiers and tax forms will be required for compensation purposes (i.e. W-9 form, SSN, V#, addresses, etc.)
- Total Monetary Amount:
- Focus Group (Part 1): Each participant in the focus group will receive a total compensation of \$150 (\$75 for each session) for their involvement in two sessions.
  - · Intervention (Part 2): Participants in the intervention group will receive \$150 for completing both the pre and postsurveys ( \$75 for each survey)
- Satisfactory Survey Compensation: Participants who complete the survey will receive \$50 as compensation.
- 2. Type of Compensation:
- The compensation will be provided as gift card after completing each research activities.
- 3. Disbursement of Compensation:
- The compensation will be disbursed to participants through their preferred method, such as a gift card (physical or ecard) . The specific method of disbursement will be communicated to participants, and arrangements will be made accordingly
- 4. Determining the Amount:
- participants, the importance of their contributions to the study, and the prevailing compensation rates for similar studies or participant involvement. These amounts aim to provide fair and reasonable compensation for participants' time and The compensation amounts were determined based on factors such as the time commitment required from
- 5. Identifiers and Tax Forms:
- In consideration of the community's concerns and challenges, we have decided to waive the requirement of providing be a significant challenge and may hinder participation in the study. Therefore, participants will not be asked to provide Social Security Numbers (SSN) or any tax-related forms. We acknowledge that obtaining SSN from participants could SSN or complete tax-related forms.
- This decision aims to prioritize the community's comfort and trust while minimizing any barriers to participation. We

will ensure that alternative methods are in place to provide compensation to participants without the need for SSN or tax forms.

- The privacy and confidentiality of participants' personal information will continue to be respected throughout the
  compensation process. Participants will be assured that their identifying information will be handled securely and used
  solely for the purpose of compensation disbursement.
- 2. If compensation will be pro-rated, explain the payment schedule.

ID: HM20024502

HM20024502 View: SF2 - Contingency Plan

### HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN

### Contingency Plan

This page will be used by the IRB in the event that an institution-wide emergency situation arises that requires contingency plans. A contingency plan describes the alternative procedures that a study would want to use in case of an emergency that approve alternative study activities along with criteria for when those activities would or would not be put into effect. prevented normal study activities from occurring. It is a form of adaptive protocol. It enables the VCU IRB to quickly For example, in 2020, some studies had a COVID-19 Contingency Protocol approved that described alternative remote procedures that they would switch to whenever the University restricted in-person research activities.

that have to be submitted to the IRB and should reduce the number of incidents of deviations and noncompliance by inclusion criteria, etc. Flexibility and adaptations that are built into the protocol will reduce the number of changes In all studies, investigators are strongly encouraged to plan prospectively and build flexibilities into their regular emergency situation. For example, windows for timed study visits, ranges instead of exact values, flexibilities in protocols (regardless of whether an emergency situation exists) as well as think about what they would do in an

Further instructions and smartform questions on this page will be released from the IRB in the event of such an institution-wide emergency situation.

7/8/23, 9:07 AM

HM20024502 ID: HM20024502

View: SF2 - Research Plan Complete

PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

### Research Complete

Protocol Progress:

- **INITIAL SETUP**
- **■** BACKGROUND, RATIONALE & GOALS
- **RESEARCH PLAN**
- (d) CONSENT PLAN (g) RISKS, PRIVACY & CONFIDENTIALITY (d) POPULATIONS WITH SPECIAL CONSIDERATIONS (7) INSTITUTIONAL REQUIREMENTS (8) DOCUMENTS

Click Continue below to go to the next section

View: SF2 - Consent Process HM20024502 ID: HM20024502 7/8/23, 9:07 AM

### methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn

### Consent Process

1. \* List all consent groups:

Roles

Waivers

Types

Group

Requested

by Participant Consent

group consent form

No Waivers

Signed

View Focus

Re-

Consent from out list if study, we will conversation after the first we have not **Coercion Decision** Two weeks participant heard back about the drop the from her. process for the beside the mandatory wait period to go home before they participant over them instead of participant Having a the Community and think after receiving standing for the Sitting /assent down Board During sign provided with a focus group or cancer among RB approval, Depending on May 2023, at about cervical the education private room oackground session, the expected in the consent either in the Roles Electronic -Other Signatures participants provided by commence Center in a he Islamic discussion, enrollment, consenting study will Advisory women. Muslim will be their platform for DocuSign (standard regulated non-FDA studies) Research Coordinator Lead Student/Trainee Principal Investigator Investigator (leading Co/Sub-Investigator Research Assistant their own project)

details of the

Waivers Roles

**Types** 

Group

Roles Electronic -Other Signatures

**Coercion Decision** 

Consent Re-

> components respective explained. will be

will provide the participant with The discussion decision about potential risks, discussion will assistant (RA) the necessary information to compensation with the study. materials and -The consent take place in-The research will cover the benefits, and participation. face-to-face allowing for interaction associated informed make an person,

DocuSign The the opportunity decision. They -Participants will be given will be offered and make an electronically the option to participation using either to consider electronic informed consent provide their

Group

| Re-<br>Consent |
|-------------------------------------------|
| <b>Coercion Decision</b> |
| Roles Electronic<br>-<br>Other Signatures |
| s Roles |
| Waivers |
| Types |

Signatures Consent Coercion Decision

consent form

will be
accessible via
a provided link,
ensuring
convenience
and ease of
use for the
participants.

-Ongoing reconfirmation of consent is not applicable in this study.

circumstances and think to two weeks) before they to make a depending on duration may will be given **Participants** to go home from a week participation n the study. regarding their he exact expecting sufficient decision time( vary and the participant mandatory wait period Having a slamic Center consent for the /assent obtained at the sign consent before opportunity to group will be **Consent Will** will have the **Participants** engaging in Consent for intervention When and during the scheduled education sessions provide Where Occur: the platform for DocuSign (standard regulated non-FDA studies) Trainee/Student(working Research Coordinator Lead Student/Trainee Principal Investigator Investigator (leading Research Assistant their own project) on project) Requested Waivers

Consent by Participant

group consent form

View Intervention Signed

much time as

encouraged

are

What Will Be

to take as

participants

they need to

Discussion:

During the

consent

During the

Consent

Covered

review the

provided

complexity of

the study.

educational

program.

Fypically,

| Ö |
|-------------------------------------------|
| Roles Electronic<br>-<br>Other Signatures |
| ctronic<br>nature |
| Roles Electronic<br>-<br>Other Signatures |
| 8.₹ |
| Roles |
| Waivers Roles |

Types

Group

Re-Consent questions, and consider their interests their decision. lime to make coercion Decision decision and preferences that there is an informed participants information, emphasize choice that are free to aligns with no rush to necessary The study team will take the make a that provided with a involvement. They will have along with any potential outcomes. The may arise from informed about topics covered, the opportunity including confidentiality program, including the questions and explanation of nature of their their rights as duration, and discomfort or will be clearly participation participants, participants educational educational Additionally, participants effects that discussion, associated explained, expected sessions voluntary risks and research session benefits adverse and the detailed will be with the

7/8/23, 9:07 AM

Waivers Roles

**Types** 

Group

Roles Electronic -Other Signatures

**Coercion Decision** 

Re-Consent

clarifications before

providing

consent.

How the Consent

Discussion Will Occur:

discussion will The consent

occur inperson,

allowing for

communication direct

research team between the and the

participants. A designated

research team member, such research as the

will conduct

assistant (RA), the discussion in a private

room at the Islamic Center.

The participant opportunity to will have the

consent form, review the ask any

questions, and before making an informed discuss any concerns

participate. The RA will be decision to

available to provide

Waivers Roles Sign

**Types** 

Group

Roles Electronic -Other

Coercion Decision

Re-Consent

explanations and guidance as needed to ensure the participant's understanding of the study and their role in it.

group will be participating in the study at any time, even after providing initial consent. on an Ongoing will ensure that reconfirmation not applicable research team withdraw from information to How Consent Reconfirmed However, the provided with of consent is are aware of their right to the research in this case reach out to participants **Participants** intervention educational team if they will also be a one-day Since the program, have any ongoing Will Be contact Basis:

questions or

| Coercion Decision |
|-------------------------------------------|
| Roles Electronic<br>-<br>Other Signatures |
| Waivers Roles |
| Types |
| Group |

Re-Consent

concerns
during or after
the
educational
program.

2. Upload any consent / assent documents:

| | Document<br>Name | Document \ | Version Date Upl<br>Modified By | <b>Date</b><br>Modified | Uploaded <sub>Type</sub><br>By | Туре | Approved |
|---|---|---|---|---|---|---|---|
| View | Consent form focus group | Namoos- Consent 0.03<br>from of focus<br>group<br>05.12.2023.pdf | | 7/8/2023<br>1:09 AM | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | Yes |
| View | Consent form -<br>Intervention<br>program | Namoos- Consent 0.04 from of Intervention group 05.12.2023 copy.pdf | · | 7/8/2023<br>1:09 AM | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | Yes |
| View | View Fund Plan | Asmaa -Budget<br>04.13.2023.xlsx | 0.03 5 | 5/12/2023<br>11:52 AM | Asmaa<br>Namoos | Funding Proposal | Not<br>Applicable |
| View | Education<br>session | Asmaa Education 0.02 session guide , intervention group-04.07.2023.docx | | 5/12/2023<br>10:52 AM | Asmaa<br>Namoos | Other | Yes |
| View | View Timeline Plan | Namoos, timeline (for PROMIS women Projectdocx | 0.02 5 | 5/12/2023<br>10:43 AM | Asmaa<br>Namoos | Other | Yes |
| View | Conceptual<br>model | Asmaa<br>Conceptual Model<br>05.12.2023.docx | 0.02 5 | 5/12/2023<br>10:40 AM | Asmaa<br>Namoos | Research Measure | Yes |
| View | View Flayer 2 | Asmaa Flyer<br>Version<br>05.12.2023.docx | 0.01 5 | 5/12/2023<br>10:39 AM | Asmaa<br>Namoos | Other | Yes |
| View | Namoos-Focus<br>group script<br>guide | Namoos -Focus<br>Group Script<br>Guide.docx | 0.02 5 | 5/12/2023<br>10:24 AM | Asmaa<br>Namoos | Other | Yes |

| | Document<br>Name | Document | Version | Version Date Up | Uploaded Type<br>By | Туре | Approved |
|---|---|---|---|---|---|---|---|
| View | Participants -RA Namoos-communication Participar script communi | Namoos-<br>Participants -RA<br>communication<br>script .docx | 0.01 | 5/12/2023<br>6:45 AM | Asmaa<br>Namoos | Other | Yes |
| View | Study Survey(<br>Pre-post and<br>satisfactory<br>scales) | Survey- Promise<br>women project<br>05.12.2023.docx | 0.01 | 5/12/2023<br>6:35 AM | Asmaa<br>Namoos | Research Measure | Yes |
| View | View consent form-<br>focus group | Consent from -<br>Focus group<br>02.20.2023.docx | 0.01 | 2/20/2023<br>4:32 PM | Asmaa<br>Namoos | Consent/Assent/Information No<br>Sheet | ON |
| View | View VS biosketch | Sheppard<br>Biosketch for AN<br>11.14.2022.pdf | 0.01 | 2/20/2023<br>4:00 PM | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |
| View | Communication<br>log | Communication log.docx | 0.01 | 2/20/2023<br>3:59 PM | Asmaa<br>Namoos | Other | Yes |
| View | View PRMC approval 2022-10-10-10-10-10-10-10-10-10-10-10-10-10- | 2022-10-<br>10_MCC-22-<br>19873_PRMC<br>Approval<br>Letter.pdf | 0.01 | 10/10/2022 Asmaa<br>12:30 PM Namoo | Asmaa<br>Namoos | Ancillary Committee<br>Approval | Not<br>Applicable |
| View | View F <b>lye</b> r | Flyer<br>004.08.2022.png | 0.01 | 4/8/2022<br>6:09 PM | Asmaa<br>Namoos | Other | Yes |
| View | Namoos<br>Resume | Dr. Namoos A.<br>Biosketch<br>06.07.2021.pdf | 0.01 | 4/3/2022<br>3:47 PM | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |

View: SF2 - Consent Plan Complete

HM20024502

ID: HM20024502 7/8/23, 9:07 AM

PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

### Consent Plan Complete

Protocol Progress:

- **INITIAL SETUP**
- **■** BACKGROUND, RATIONALE & GOALS
- RESEARCH PLAN
  - **CONSENT PLAN**
- ⑤ RISKS, PRIVACY & CONFIDENTIALITY⑥ POPULATIONS WITH SPECIAL CONSIDERATIONS
  - (7) INSTITUTIONAL REQUIREMENTS (8) DOCUMENTS

Click Continue below to go to the next section

ID: HM20024502 HM20024502

View: SF2 - Risks, Discomforts, Potential Harms and Monitoring

### HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN

## Risks, Discomforts, Potential Harms and Monitoring

- 1. \* Describe the risks of each research procedure to participants or others. For each identified risk, provide an assessment of the anticipated seriousness and likelihood of the risk. Some examples of possible risks include but are not limited to:
- Physical risks (e.g. bodily harms or discomforts, side effects, etc.)
- Psychological risks (e.g. emotional, mental, or spiritual harms or discomforts, changes to thoughts, beliefs, or behaviors, etc.)
- Research data risks (e.g. loss of confidentiality and privacy)
- Social or legal risks (e.g. impacts on relationships or reputation, legal or criminal justice actions for self or others, etc.)
- Financial risks (e.g. impacts on income, employability, or insurability, loss of services, etc.)
- Other risks (e.g. unforeseeable risks of experimental procedures, risks related to particular study designs (randomization, washout, placebo, withholding care/services, deception), etc.)

See the help text for additional guidance.

Physical risks: NA

esearch study. The research team is committed to maintaining confidentiality and ensuring the highest level of data nherently involves some level of privacy loss. Although stringent measures will be in place to protect your personal Psychological risks: Participation in the study may entail psychological risks, as some of the questions asked may information, there is a small risk of unauthorized access or misuse of your data by individuals not involved in the potentially cause discomfort or evoke emotional responses. It is important to note that participating in research security to minimize such risks.

potentially access and misuse your personal information. Additionally, there is a possibility of confidentiality breaches during the transfer and storage of research data. The research team is committed to implementing rigorous security Research data risks: Participating in this research study may involve some degree of privacy loss. It is important to acknowledge that there is a small inherent risk that unauthorized individuals outside of the research study could measures to minimize these risks and ensure the confidentiality and integrity of your data.

Social or legal risks: Participation in this study may involve social or legal risks related to cultural sensitivity. It is mportant to recognize and respect the diverse cultural backgrounds of participants and their communities. The

research team acknowledges the need to seamlessly interact with individuals from different cultures by understanding and adhering to the norms, customs, and values of each specific culture.

provide training to researchers to enhance their cultural competence and sensitivity when working with participants interactions are culturally appropriate and considerate. The team will make efforts to establish clear guidelines and By promoting cultural sensitivity, the research team aims to create an inclusive and respectful environment for all participants. This involves taking proactive measures to ensure that research procedures, communication, and rom various cultural backgrounds.

social or legal risks that may arise due to cultural misunderstandings or insensitivity. This will help facilitate effective communication, build trust, and create an atmosphere where participants feel comfortable and respected in sharing By fostering a culturally sensitive approach throughout the study, the research team aims to minimize any potential their experiences and perspectives.

Financial risks: NA

## 2. \* Describe how each of the risks/harms/discomforts identified above will be minimized:

mplemented. Participants will have the option to take breaks during the study if needed, ensuring their well-being and committed to ensuring that participants' mental health and emotional well-being are prioritized throughout the study. esources and information about counseling services, should they require additional support. The research team is Psychological Risks: To minimize psychological risks and address emotional discomfort, several measures will be allowing them to manage any emotional distress that may arise. Additionally, participants will be provided with

implemented. De-identification and coding processes will be employed to remove any identifying information from the data, ensuring confidentiality. The interview answers will be recorded using an electronic data capture system hosted on secure VCU servers accessible only to authorized researchers. These servers comply with stringent security Research Data Risks: To mitigate research data risks and ensure participant privacy, robust measures will be protocols and maintain researcher-only access, further safeguarding the confidentiality of participant data

and alignment with cultural norms. Community leaders from the target population will provide input and review religious study is a member of the same community and has prior experience conducting studies in Islamic centers, establishing Social or Legal Risks: To address social or legal risks, several strategies will be employed to ensure cultural sensitivity researcher, creating a safe and comfortable environment for participants. The education sessions will be conducted in and community engagement. Expert researchers will review the educational sessions to ensure their appropriateness frust and rapport. The research team will consist of female members only, including the peer researcher and primary materials included in the sessions, ensuring cultural accuracy and relevance. The research assistant involved in the a private setting within the mosque, respecting the cultural and religious values of the participants and maintaining

## 3. \* Describe any potential risks or harms to a community or a specific population based on study findings (e.g. information that could be stigmatizing or derogatory):

be sought through the guidance of the Imam, who will introduce the research to the community. The research team has here is no identified community risk associated with the study findings. The community's acceptance and support will The project will be conducted within the Islamic centers among a conservative community. It is important to note that an established project with the community and maintains a community bridge, fostering trust and collaboration.

accurate, and align with the values and norms of the community. The involvement of the CAB adds an additional layer To ensure cultural sensitivity and appropriateness, the study material will undergo review by the Community Advisory Board (CAB). This review process will help ensure that the study findings, information, and materials are respectful of protection against any stigmatizing or derogatory information.

By actively engaging with the community, seeking guidance from community leaders, and involving the CAB, the study

https://irb.research.vcu.edu/irb/app/portal/smartform/printProject/\_Protocol/7B0E8344A95711ECC991CBE9AD565000?packetIds=defaultPrintPacket

aims to minimize any potential risks or harms that may arise from the dissemination of study findings. The overall goal is to promote understanding, respect, and positive engagement within the community and to ensure that the study findings contribute to the well-being and empowerment of the target population.

### 4. Where appropriate, discuss provisions for ensuring necessary medical, professional, or psychological intervention in the event of adverse events to the subjects:

Provisions for ensuring necessary medical, professional, or psychological intervention in the event of adverse events to he subjects will not be applicable in this study. Since there are no anticipated medical, professional, or psychological expected. However, if any unforeseen adverse events were to occur during the study, the research team would take isks associated with the study, the need for intervention or support services in response to adverse events is not appropriate measures to address them promptly and ensure the well-being and safety of the participants.

## $5.~^\circ$ Describe criteria for when the investigator would withdraw an individual participant from the study; such as safety or toxicity concerns, emotional distress, inability to comply with the protocol, etc.:

The investigator may withdraw an individual participant from the study based on various criteria, including but not imited to: Safety Concerns: If the participant experiences any adverse effects or safety concerns related to the study procedures, interventions, or materials, the investigator may consider withdrawing the participant to ensure their well-being and

overwhelmed, or difficulty relaxing, the research assistant (RA) will be attentive and responsive. The RA will provide support and, if necessary, stop the conversation in a considerate manner. The participant will be given the choice to Emotional Distress: If the participant exhibits signs of emotional distress, such as symptoms of anxiety, feeling continue or discontinue the conversation, respecting their emotional well-being.

consider withdrawing the participant. This ensures that the study remains valid and maintains the integrity of the data Inability to Comply with the Protocol: If the participant faces challenges in complying with the study protocol, such as difficulty attending scheduled sessions, completing required tasks, or following instructions, the investigator may

eview the participant's case and make a decision on whether to continue their participation or withdraw them from the consequences. If the participant chooses to continue despite experiencing emotional distress, the RA will resume the It is important to note that the participant will be informed of their right to withdraw from the study at any time without conversation to prevent any potential embarrassment. The PI will be notified of the situation, and the study team will study, taking into consideration their well-being and the study's objectives.

## 6. \* Summarize any pre-specified criteria that would trigger the investigator/sponsor/monitoring committee to stop or change the study protocol due to safety concerns:

covid 19 crisis, the study could stop/hold due to the pandemic. This will be done according to the research workflow at The research team follows the VCU policy regarding safety concerns. Since we are in a critical time of year due to the

### Data and Safety Monitoring

Data and safety monitoring is a system for checking the study's data at regular intervals over the study period to identify and address issues that could affect the safety of research participants. This requirement is in accordance with 45 CFR 46 111

The purpose of data and safety monitoring plan is to set forth study team procedures for monitoring/addressing:

- Participant safety (physical, psychological, etc.)
- Data validity
- Early stopping (termination) based upon changes in risks and benefits.

7. \* Indicate if this study will have a Data Safety Monitoring Board (DSMB) or a Data Safety Monitoring Plan (DSMP): [Required for all greater than minimal risk studies]

HM20024502 View: SF2 - Privacy

ID: HM20024502

### PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

#### Privacy

Privacy refers to an individual's right to control how others view, record, or obtain information about them. When privacy is violated it can involve such things as

- Being asked personal questions in a public setting;
- Being publicly identified as having a particular characteristic or diagnosis;
- Being seen entering a place that might be stigmatizing;
- Being photographed, videotaped or observed without consent;
  - Disclosure of personal information to unauthorized people

Privacy is not the same as confidentiality because privacy protections apply to people, and confidentiality protections apply to data. Confidentiality protections should be described on the Data Confidentiality page of this form, not here.

#### Instructions for this page:

study. The options listed include some of the most common best practices. Not all will be applicable to every study. Select all the applicable ways that the research team will protect participants' privacy throughout the course of the

\*\*The IRB will expect studies to operationalize all selected checkboxes into the conduct of the research

To elaborate on any response, also click the "Other Protections" checkbox to provide further explanation in the last free-text question.

Read the entire page before filling out the form.

- 1. \* Protections when conducting one-on-one in-person interventions or interactions (for groups see Q2 below):
- Conducting study activities in locations that maximize privacy (limited people around, closing doors, drawing drapes around beds, monitoring voice volume, etc.) >
- Verifying identity before discussing personal information.
- Asking the participant if they are comfortable answering questions in that location
- Asking the participant if they are comfortable with having other people present (if any)
- Moving away from other people when conducting activities in public spaces or offering a private space

Using generic signs on research rooms and spaces, particularly for research on stigmatizing or sensitive topics Using generic signs on research rooms and spaces, particularly for research on stigmatizing or sensitive topics Collecting paper forms in a closed box or envelope rather than passing to others or leaving in an open Asking everyone in a public group setting (e.g. classrooms, workshops) to turn something in (blank or Limiting participant identifiers that would be visible on paper documents (i.e. using study IDs instead Offering other options of ways to respond to sensitive questions (i.e. pointing, clicking, or writing) if Offering other options of ways to respond to sensitive questions (i.e. pointing, clicking, or writing instead of Discussing privacy with the participants and the importance of not talking outside the group about Conducting study activities in locations that maximize privacy (limited people passing by, closing Allowing participants to use a pseudonym or limiting use of individuals' names during the group Allowing people to distance themselves from other participants during group activities Ensuring non-participating individuals are not captured on recordings or in photos filled) so participants do not have to self-identify when turning in materials Moving to a more private area to answer questions or to discuss concerns N/A - study has no in-person interventions or interactions with participants 2. \* Protections when conducting group interventions or interactions: Other protections not listed in this question – describe below Other protections not listed in this question – describe below N/A - study has no group interventions or interactions what other people say during the group session doors, monitoring voice volume, etc.) uncomfortable verbally responding of direct identifiers) speaking) activity >

3. \* Protections when conducting remote interventions or interactions (e.g. phone, text, email, video-conference, tele-health, online, etc.):

| Conducting study activities in locations where study staff can maximize their own privacy (limited people around, closing doors, monitoring voice volume, etc.) |
|---|
| Leaving/sending generic messages that avoid using study and participant identifiers, such as names, study titles, clinics, study topics, etc. |
| Obtaining permission prior to sending text messages |
| Advising the participant to move to a location where they are comfortable answering questions and will not be overheard - incorporate this instruction into your study materials |
| Advising online participants to complete the activity at a time and location where they will be comfortable answering questions - incorporate this instruction into your study materials |
| Ensuring non-participating individuals are not captured on recordings or in photos |
| Offering other options of ways to complete the activity (i.e. online, paper, phone) if more privacy is desired |
| Offering a way to save and return later to the online activity if privacy is compromised |
| Other protections not listed in this question — describe below |
| N/A – study has no remote interventions or interactions with participants |

- 4. \* Protections when mailing study materials to/from participants:
- Obtaining permission to mail study materials
- Confirming/verifying the accuracy of addresses before mailing items
- Ensuring the participant is able to personally receive mailed materials and has a way to protect their own privacy if they do not want others to know they are receiving research communications (i.e. notifying participants of when to expect it) >
- Using return address labels and document headers that avoid study identifiers, such as study names, clinics, study topics, etc.
- Avoiding or limiting use of participant identifiers and health information on mailed documents (i.e. using study IDs instead of direct identifiers)
- Providing a return mailing address label or pre-addressed envelope to ensure returned items are sent to the correct address
- Communicating receipt of mail from participants and/or asking them to notify you when they mail it to ensure study documents are not lost in transfer
- Offering other options of ways to complete the activity (i.e. by phone or online) if desired

6. Describe any other way(s) that the research team will protect participants' privacy. See the help text for additional guidance.

During our intervention we will take pictures after verbal approval from the ladies who are in the room, for more protection we will blurred the faces and use these pictures during conference only. View: SF2 - Data Confidentiality and Storage

HM20024502

HM20024502

ID: HM20024502

7/8/23, 9:07 AM

methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn

## Data Confidentiality and Storage

maintained and shared. It describes how the study's research materials (data, specimens, records, etc.) are protected Confidentiality refers to the way private, identifiable information about a participant or defined community is from unauthorized access.

| | ٠ | i |
|---|---|---|
| | a | |
| | ř | |
| | 2 | |
| | a | |
| | 9 | |
| | a | |
| | Ľ | |
| | c | |
| 1 | Ŧ | |
| | Ĺ | |
| | 7 | |
| ٠ | 2 | |
| | • | |
| | u | į |
| | c | |
| | 7 | ١ |
| | 2 | |
| - | F | |
| | c | ١ |
| | Ξ | |
| | Ξ | |
| , | ٠ | |
| | u | į |
| | c | |
| ٠ | Ξ | |

Select all the ways that the research team will keep the study materials and data confidential throughout the course of the study. Not all will be applicable to every study.

To elaborate on any response, also click the "Other Protections" checkbox to provide further explanation in the last free-text question.

### Read the entire page before filling out the form.

| materials: |
|-------------|
| research |
| paper |
| for |
| Protections |
| * <u>-</u> |

| | ( | ) |
|---|--------|-------------|
| | Captro | 5 |
| | | Manicalling |
| | 1 | > |
| _ | | |

| nen at an off-campus location |
|-------------------------------|
| ₹ |
| including |
| at all times, |
| 를 |
| at |
| documents |
| ē |
| ap |
| of p |
| control |
| Maintaining |

| 0 | |
|------------------------|-------|
| tead | |
| ins | |
| ly IDs in | |
| ρŗ | |
| ) sti | |
| sing st | |
| ents (i.e. usi | |
| s (i. | |
| ent | |
| uno | |
| er document | |
| aper | |
| tifiers on paper docun | |
| rs o | |
| tifie | |
| den | |
| änti | |
| Sign | |
| arti | |
| e of particip | |
| nse | |
| ing | |
| voiding us | ers) |
| | ntifi |
| iting or avoid | de |
| niti | ect |
| Ē | € |
| | _ |

| personnel |
|------------|
| study |
| horized |
| ly to autl |
| sible only |
| accessible |
| locatior |
| secure |
| i. |
| documents |
| ng paper |
| Storin |
| > |

| Promptly transcribing, scan | nning, c | lbing, scanning, or abstracting da | data | data from paper into el | into | electronic | platforms w | vith |
|---|---|---|---|---|---|---|---|---|
| destruction of the paper copy | ۸dc | | | | | | | |

| cords (and obtaining prior permission when required) in accordance | |
|---|---|
| hen require | |
| permission w | |
| btaining prior | |
| f paper records (and o | nt policies |
| Proper destruction of paper recor | with VCU Records Manageme |
| Prope | with \ |

| describe below | |
|---|---|
| n not listed in this question – describe belo | naterials |
| rection not listed | N/A – no paper research materia |
| Otner protectio | N/A – no p |
| | L |

### 2. \* Protections for research specimens:

| 5 |
|----------------------------------------------------------------------|
| ocati |
| sndu |
| I-call |
| an o |
| en at |
| m gr |
| cindir |
| es, ⊟ |
| เรลเ |
| l ot specimens at all times, including when at an on-campus location |
| spe<br>spe |
| s to loninos gr |
| g<br>S |
| IIall |
| Mal |

| (I) |
|----------|
| Ĕ |
| 5 |
| Š |
| ē |
| Q |
| ⋛ |
| ĭ |
| stn |
| О |
| ě |
| ĽŽ |
| 2 |
| ŧ |
| æ |
| 5 |
| ⋛ |
| on |
| a) |
| sible |
| : |
| S |
| cce |
| ŏ |
| ğ |
| 5 |
| ä |
| 8 |
| <u>ŏ</u> |
| a) |
| Ξ |
| ರ |
| Se |
| œ, |
| č |
| .= |
| S |
| ē |
| Ε |
| .⊡ |
| e |
| ş |
| б |
| .⊑ |
| ö |
| 윥 |
| 5, |

| , o.o. , | 7007707 |
|---|---|
| | When providing devices or mobile apps to children, informing parents about the settings and how to manage them (if applicable), internet access, and any other installed apps on the device |
| | Other protection not listed in this question – describe the device/app and protection below |
| > | N/A – no computers or devices/apps being provided for participant use outside the lab |
| 5 * Pro | Protections for email/online communications |
| > | Only using VCU/VCU Health email addresses for study-related communications |
| > | Only using VCU/VCU Health–approved methods of teleconferencing or video conferencing (e.g. Zoom)<br>(for studies involving HIPAA, contact VCU or VCU Health Information Security [as appropriate] about<br>HIPAA-compliant systems) |
| | Other protection not listed in this question — describe below |
| | N/A – no email/online communications |
| 6. Spec<br>be st | Specify any other places where this study's paper and electronic research data and/or physical specimens will<br>be stored and any other ways they will be secured from improper use and disclosure. |
| See t<br>NA | See the help text for additional guidance.<br>NA |
| 7. * If re the P the P 1) ide organ organ 2) giv | * If research data/specimens will be sent/released to person(s) or group(s) outside of the VCU study team or the PI's department for the conduct of this protocol (not for future sharing), 1) identify the data/specimen recipient(s) along with their VCU department or other institutional or organizational affiliation(s). 2) give a description of what identifiers and/or codes will accompany the data/specimens. If data/specimens are not being sent/released outside of the VCU study team or the PI's department, state that: |
| 8. * Sele<br>gathe | * Select all identifiers that will be collected <u>at any time</u> as part of this study (including for recruitment, data<br>gathering, data analysis, etc.), even if the data will eventually be anonymized: |
| <b>&gt;</b> | Names |
| > | Geographic Locators Below State Level |
| | Social Security Numbers |
| | Dates (year alone is not an identifier) |
| | Ages over 89 (age under 89 is not an identifier) |
| > | Phone Numbers |

9. \* If the study will code (i.e. de-identify) the research data by replacing subjects' names and/or other identifiers with assigned subject IDs, explain the following aspects of the coding process:

No Identifiers

Employee V#

- The process for how subject IDs will be generated/assigned (e.g. random, sequential) - Whether there will be a key that links the subject ID with direct identifiers. If there will be no linkage key, state

If a key will be created, describe

- The place where the key will be stored

- The role(s) of all individuals who will have access to the key

-When the key will be destroyed

See the help text for guidance.

In this study, the research data will be coded by replacing participants' names and other identifiers with assigned subject IDs to ensure confidentiality and protect privacy. The coding process will follow the following aspects:

participant will be assigned a unique identifier that is unrelated to their personal information or characteristics. This Generation/Assignment of Subject IDs: Subject IDs will be generated using a random assignment process. random assignment helps maintain anonymity and protects the participants' identities.

subject IDs. However, in this study, there will be no linkage key that links the subject ID back to direct identifiers. The Linkage Key and Storage: A linkage key will be created to associate the original patient identifiers with the assigned coding process ensures that the data remains de-identified and confidential.

database. Only the Principal Investigator (PI) would have access to the linkage key. The PI would be responsible for Storage of the Linkage Key: If a linkage key were created, it would be stored separately in the secure REDCap safeguarding the confidentiality of the key and ensuring that access is restricted to authorized individuals.

individuals involved in the study would have access to the linkage key to further ensure the security and privacy of the Access to the Linkage Key: The PI would be the sole individual with access to the linkage key. This access is granted to ensure the integrity of the coding process and to maintain the confidentiality of the participants' data. No other participants' information.

Destruction of the Linkage Key: Once the study is completed, the original identifiers and linkage keys will be securely destroyed. This step ensures that any potential re-identification of participants' data is prevented, further protecting heir privacy and confidentiality. By employing these coding procedures and secure storage practices, the study ensures that participants' data remains de-identified and confidential throughout the research process.

View: SF2 - Data Retention

HM20024502

ID: HM20024502

7/8/23, 9:07 AM

HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn

### Data

4. \* Will audio/video recordings and full face photographs be destroyed?

Other

ON (

Yes

5. If yes, describe at what point and how recordings will be destroyed: They will be destroyed at the end of the study

6. If no, explain why the recordings need to be maintained:

View: SF2 - Sharing Plan HM20024502

ID: HM20024502

### PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

#### Sharing Plan

This page addresses times when investigators may be required to share information about participants or may desire to share their research information/specimens with the aim of advancing science. This page creates a plan for when and how information/specimens could be shared.

Try to anticipate all reasonably foreseeable sharing so that the consent document can also reflect that information. However, it is acceptable to amend this page later and explain either how re-consent of previously and currently enrolled participants will occur or why re-consent should not be required.

Respect for Persons by confirming that plans for sharing do not go against what participants would understand The IRB reviews this page against the consent document (if one exists) to demonstrate the ethical principle of about the use of their data/specimens.

The IRB also ensures there are adequate protections for the privacy of participants and the confidentiality of participants' data/specimens when data is shared with others. 1. \* Is it likely investigators could discover information about child/elder abuse or neglect that would require mandatory reporting by the investigators or staff?

The Code of Virginia requires that most medical personnel and all employees of institutions of higher education report suspected child/elder abuse or neglect.



ŝ

2. \* Is it likely investigators could discover a previously unknown reportable disease or condition that would require mandatory reporting by the investigators or staff (i.e., HIV, coronavirus, hepatitis, etc.)?



ŝ

3. \* Will the sponsor or investigator obtain a Certificate of Confidentiality for this study?

Certificates of Confidentiality (CoC) are issued by the National Institutes of Health (NIH), the FDA and CDC to regardless of funding can qualify to receive a CoC. A CoC is automatically issued for research that was protect identifiable research information from forced disclosure. All human subject research studies ongoing on December 13, 2016, or initiated after that date. For more information, see ttps://humansubjects.nih.gov/coc/

Yes - CoC has been obtained or issued automatically

No - Will not obtain CoC for this study

7/8/23, 9:07 AM

| Will not use information/specimens for purposes beyond this study. | ✓ Not sure and will submit an amendment when known | Other use(s) of individual-level information in a way not listed above | <ol> <li>* Select the way(s) the VCU PI/study team may share information or biospecimens (including DNA) with other researchers who are not on this study team (i.e. for analyses beyond/apart from the aims of this study).</li> <li>See help text for definitions.</li> </ol> | Will share directly identifiable information or specimens with other researchers. | ('Directly identifiable' means that identifiers like name, medical record number, social security number, etc. are included in/attached to the dataset/specimens. Maintaining identifiable data for future research uses is treated by the VCU IRB as a registry. The data recipient's use of identifiable data would require them to obtain IRB review. VCU IRB studies will be asked more questions about this on a later page.) | Will share de-identified or indirectly identifiable information or specimens with other researchers. | ('De-identified' means that a linkage/Rey code exists that links identifiers to data/specimens. The VCU researcher maintains the key but does not share it with any other researchers. The recipient's use of de-identified data/specimens may not be human subject research if there is documentation that the key will never be shared with the recipient, but they should check with their own IRB about review requirements. VCU IRB studies will be asked more questions about this on a later page.) | Will share anonymized information or specimens with other researchers. | ('Anonymized' means that 1) no linkage/key codes exist that link identifiers to data/specimens; and 2) subjects cannot be readily identified (i.e. no direct or indirect identifiers or identifiable combinations of variables). The VCU IRB considers uses of anonymized data/specimens by other researchers to not be human subject research, but the recipient should check with their own IRB about review requirements.) | Will only share aggregate results (summary-level results), not individual-level information or specimens. | (The VCU IRB considers uses of aggregate data to not be human subject research because there are no individual subjects. The data recipient should check with their own IRB about review requirements.) | Will contribute to an existing registry or repository (VCU IRB studies will be asked more questions about this on a later page.) | Will submit data to an NIH genomic data repository (VCU IRB studies will be asked more questions about this |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

| Will not share information/specimens with other researchers. | Not sure and will submit an amendment when known | Other sharing of individual-level information with other researchers | <ul> <li>Since you responded in a question above that you may use or share anonymous, individual level data, indicate why the proposed use or sharing of anonymous data/specimens is not inconsistent with what participants would have reasonably understood from the consent document about the uses of their information. (Select all that apply.)</li> </ul> | The consent form states that after identifiers are removed, information or specimens could be used for future research studies without additional informed consent from the subject (this is a new element of consent included in consent templates as of May 2018) | The consent form or exempt information sheet is silent about whether/how information or specimens could be used for future research studies. | The information or specimens were/will be obtained under a waiver of informed consent, waiver of HIPAA authorization, or an exempt study that did not use an information sheet. | Other reason why anonymous use/sharing is not inconsistent with the consent document |
|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|

- 7. \* The Principal Investigator certifies that prior to releasing an anonymized dataset or anonymized specimens the following conditions will all be met:
- all 18 HIPAA identifiers (including all dates) will be removed;
- all indirectly identifiable data elements (unusual, rare, uncommon data) will be removed, grouped, suppressed, or otherwise transformed to no longer be readily identifiable;
- a different subject ID will be assigned than the one used for the main study and a linkage key will not be
- the PI will review the dataset/specimens to confirm that the remaining information could not be used alone or in combination with any other information to re-identify the participants represented in the data

See help text for more information.



<sup>8</sup>

- conditions will be met whenever individual level research information and/or specimens are used or shared: 8. \* The Principal Investigator certifies that after the study has been closed with the VCU IRB, the following
- The identities of participants who are represented in the dataset/specimens will not be readily ascertainable or otherwise re-identifiable by the recipient;
  - If a linkage/code key is created, it will be maintained at VCU and not shared with the recipient under any circumstances
- The PI will have no knowledge that the remaining information could be used alone or in combination with

HM20024502 7/8/23, 9:07 AM

any other information to identify the individuals represented in the data; and - The PI agrees to abide by this sharing plan even after the study has been closed with the VCU IRB.

Yes

§ O

N/A - No sharing will occur

| . If the | e Certificate of C | . If the Certificate of Confidentiality has been obtained by the PI, upload it here: | oeen obta | ined by the | PI, upload | it here: | |
|---|---|---|---|---|---|---|---|
| | Document<br>Name | Document | Version | Date Up<br>Version Modified By | Uploaded <sub>Type</sub><br>By | Туре | Approved |
| View | Consent form focus group | Namoos- Consent 0.03<br>from of focus<br>group<br>05.12.2023.pdf | 0.03 | 7/8/2023<br>1:09 AM | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | . Yes |
| View | Consent form -<br>Intervention<br>program | Namoos- Consent 0.04 from of Intervention group 05.12.2023 copy.pdf | 0.04 | 7/8/2023<br>1:09 AM | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | Yes |
| View | View Fund Plan | Asmaa -Budget<br>04.13.2023.xlsx | 0.03 | 5/12/2023<br>11:52 AM | Asmaa<br>Namoos | Funding Proposal | Not<br>Applicable |
| View | View Education session | Asmaa Education 0.02 session guide, intervention group-04.07.2023.docx | 0.02 | 5/12/2023<br>10:52 AM | Asmaa<br>Namoos | Other | Yes |
| View | View Timeline Plan | Namoos, timeline 0.02 for PROMIS women Projectdocx | 0.02 | 5/12/2023<br>10:43 AM | Asmaa<br>Namoos | Other | Yes |
| View | View Conceptual<br>model | Asmaa<br>Conceptual Model<br>05.12.2023.docx | 0.02 | 5/12/2023<br>10:40 AM | Asmaa<br>Namoos | Research Measure | Yes |
| View | View Flayer 2 | Asmaa Flyer<br>Version<br>05.12.2023.docx | 0.01 | 5/12/2023<br>10:39 AM | Asmaa<br>Namoos | Other | Yes |
HM20024502 ID: HM20024502

View: SF2 - Pertinent Results and Incidental Findings

PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn HM20024502 - Vanessa Lavene Sheppard methods among Muslim Americans WOMEN

# Pertinent Results and Incidental Findings

1. \* Is it likely investigators could discover a participant's previously unknown condition (e.g. pregnancy, disease, suicidal thoughts, wrong paternity, genetic results, or other findings that may be of importance to health or well-being) or if a participant is engaging in illegal or reportable activities:

Yes

ŝ

View: SF2 - Risk Benefit Complete

HM20024502

ID: HM20024502

7/8/23, 9:07 AM

PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

### Risk Benefit Complete

Protocol Progress:

- **INITIAL SETUP**
- **■** BACKGROUND, RATIONALE & GOALS
- **RESEARCH PLAN**
- **CONSENT PLAN**
- RISKS, PRIVACY & CONFIDENTIALITY

  ⑥ POPULATIONS WITH SPECIAL CONSIDERATIONS

  ⑦ INSTITUTIONAL REQUIREMENTS

  ⑧ DOCUMENTS

Click Continue below to go to the next section

ID: HM20024502

View: SF2 - Populations with Special Considerations

PROMIS WOMAN Education Program: ImProving ceRvical cancer prevention HM20024502 - Vanessa Lavene Sheppard methods among Muslim Americans WOMEN

### Pop

| Sulations with Special Considerations * Check all participant groups that will be either a) Specifically included in this study or b) Discernable in the research data/specimens. | |
|---|---|
| (Selections will branch) Children | |
| Emancipated minors | |
| Wards of the State | |
| Pregnant women or fetuses | |
| Neonates or Post-delivery Materials | |
| Prisoners | |
| Decisionally Impaired Adults | |
| VCU / VCUHS students or trainees | |
| VCU / VCU Health System employees | |
| Individuals with limited English proficiency | |
| Active military personnel | |
| Student populations in K-12 educational settings or other learning environments | ints |

Members of a federally recognized American Indian and Alaska Native tribe None of the Above

HM20024502 ID: HM20024502 7/8/23, 9:07 AM

View: SF2 - Populations with Special Considerations Section Complete

### HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN

# Populations with Special Considerations Section Complete

Protocol Progress:

- **INITIAL SETUP**
- **BACKGROUND, RATIONALE & GOALS**
- **RESEARCH PLAN**
- **CONSENT PLAN**
- RISKS, PRIVACY & CONFIDENTIALITY
- POPULATIONS WITH SPECIAL CONSIDERATIONS
  - (7) INSTITUTIONAL REQUIREMENTS(8) DOCUMENTS

Click Continue below to go to the next section

ID: HM20024502

View: SF2 - Study Funding

### PROMIS WOMAN Education Program: ImProving ceRvical cancer prevention methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

| တ |
|--------------|
| <b>~</b> |
| .= |
| $\nabla$ |
| $\sim$ |
| = |
| Ш |
| _ |
| > |
| $\nabla$ |
| $\bar{\neg}$ |
| # |
| ĺ |

| ÷ | |
|---|---|
| 1. Наус | 1. Have you applied for funding: Yes |
| 0 | ON ( |
| 2. Is this | 2. Is this study already funded: |
| 3. * Sele | 3. * Select all funding sources for this study (pending or awarded): |
| | Industry |
| > | Direct Federal |
| | Indirect Federal |
| | State/Local Government |
| | Non-Profit - Sponsored Project |
| | Non-Profit - Gift |
| | Internal Grant |
| | Investigator/Departmental Funds |
| | None |
| | Other |

4. \* In addition to providing funding support, what is the funding source's role in this study? Select all that apply: Collaborator in the research (helps design and/or conduct the study) [list the funder as a site on the Types of Providing guidance to the researcher but does NOT make decisions about study design Data or sample analysis regardless of identifiability Providing resources (e.g. study drug, device) Study design/Creation of the study protocol Solely providing funding support Sites page]

5. Select all related funding proposals and contracts that have been submitted through the Division of Sponsored Programs (DSP):

| RAMS-SPOT ID#<br>(FP/PT/PD#) | RAMS-SPOT ID# Direct Sponsor (FP/PT/PD#) | <u> </u> | Title | Status | StartEnd |
|---|---|---|---|---|---|
| FP00018540 | University of Kentucky Asmaa Namoos | Asmaa<br>Namoos | PROMIS Women Project | Agreement<br>Received for<br>Negotiation | |
| FP00019256 | National Cancer<br>Institute/NIH/DHHS | Asmaa<br>Namoos | Promote Cervical Cancer Proposal Under<br>Prevention Methods among Sponsor Review<br>Muslim Women in Virginia | Proposal Under<br>Sponsor Review | |

- 6. If the following conditions are ALL met, provide the index code where the HRPP will charge Single IRB (sIRB) fees associated with this review:
  - 1. The study is externally funded (fees do not apply if the study is not funded), AND
- 2. Multiple sites are executing the same research protocol (i.e. multicenter research), AND
  - 3. VCU IRB will provide IRB review on behalf of one or more non-VCU sites
- 7. \* Does the funder require the IRB to review this proposal for grant congruence?

| | • | ^ | - |
|---|---|---|---|
| ( | | | |

ID: HM20024502

View: SF2 - Types of Sites

### PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

| U | ) |
|----------------|----------|
| ±<br>U | <u> </u> |
| ) <del> </del> | -<br>> |
| U | ) |
| 0 | ) |
| - | > |

VCU Site Information

Non-VCU sites should be selected whenever any of the following situations apply:

- including being involved in the study interpretation or analysis of data and/or authorship of presentations or a) Non-VCU sites that will be collaborating on a VCU-led study (i.e. involved in conducting the research, manuscripts related to the research.)
  - b) Non-VCU sites that will be deferring to the VCU IRB for IRB review
- c) Non-VCU sites where VCU investigators will be overseeing study interventions or interactions d) Non-VCU sites/locations where VCU investigators will conduct study activities
- 2. \* Select any of the following non-VCU sites utilized in this study:

| | McGuire VAMC |
|---|---------------------|
| | Foreign Sites |
| > | Other Non-VCU Sites |

3. \* Is this a multi-center study being led by VCU?

No Non-VCU Sites

| 8<br>N |
|--------|
| Yes |
| C |

4. \* List all Non-VCU sites and locations:

Provide information only for sites that have agreed to participate or given permission for study activities to IRB, ar occur

View

| ide inform<br>ir. For Sing<br>and in thei | ation only for sites that have<br>le IRB studies where VCU w<br>ir Role indicate that site-spe | nde information only for sites that have agreed to participate or given permission for study activities to r. For Single IRB studies where VCU will be the IRB of record, list all anticipated sites that will rely on VCU and in their Role indicate that site-specific materials and agreements will be submitted in amendments. | ermission for stud<br>ticipated sites tha<br>III be submitted ir | ay activities to<br>at will rely on VCU<br>n amendments. |
|---|---|---|---|---|
| Name | Role | Adequacy | IRB FW | FWA Consultant(s) |
| The<br>University<br>of<br>Kentucky | The The University of Kentucky University (UK) collaborates with VCU investigators by actively Kentucky participating in research studies. Their role may observing the recruitment process and contributing to manuscript writing. They are not solely a location for VCU investigators but actively engage in various research activities. | In the context of research conducted at VCU collaboration with the University of Kentucky (UK), human participant safety will be observed by VCU and overseen by their Institutional Review Board (IRB). VCU, as the responsible institution, ensures that appropriate measures are in place to protect the safety and well-being of participants in the event of an unanticipated | Site<br>Engaged<br>Requests to<br>Rely on<br>VCU IRB<br>Review | |
| | | The VCU IRB provides oversight and guidance to ensure that all necessary precautions are taken to safeguard the participants | | |

5. \* How will communication occur between sites for discussion of study conduct, unexpected problems, project modifications, and interim results:

throughout the research process.

Consider the following in your response:

- how frequently communication will occur between sites

- how are sites instructed to report unanticipated problems, adverse events, or noncompliance
  - how sites can communicate needed revisions to study procedures
    - who will disseminate IRB decisions

- who will notify the IRB of potential problems and changes to the protocol

Frequency of Communication:

-Regular communication should occur between sites ( Islamic centers) to ensure coordination and address any issues that arise during the study.

-Weekly or bi-weekly conference calls or virtual meetings can be scheduled to discuss ongoing study activities progress, and any concerns or modifications required

Reporting Unanticipated Problems, Adverse Events, or Noncompliance:

-Sites should be instructed to promptly report any unanticipated problems, adverse events, or instances of noncompliance to the designated study coordinator or principal investigator.

-A reporting mechanism, such as an electronic reporting system or a designated email address, should be established to ensure efficient communication and documentation of such events.

Communicating Revisions to Study Procedures:

If sites identify the need for revisions to study procedures, they should communicate these changes to the study coordinator or principal investigator. This can be done through written reports or by submitting a formal request outlining the proposed modifications along with supporting justifications.

The study coordinator or principal investigator will review these proposed revisions and decide whether they are appropriate and feasible. If approved, the revised procedures will be communicated back to all sites.

#### Dissemination of IRB Decisions:

The Institutional Review Board (IRB) decisions, such as approvals, modifications, or disapprovals, will be disseminated by the study coordinator or principal investigator

The study coordinator or principal investigator will ensure that all relevant sites are informed of the IRB decisions in a imely manner This can be done through official written communication, email, or a secure online portal where study documents and updates are shared.

Notifying the IRB of Potential Problems and Changes to the Protocol:

It is the responsibility of the study coordinator or principal investigator to notify the IRB of any potential problems or significant changes to the study protocol.

This includes reporting adverse events, noncompliance issues, or any modifications that may impact participant safety or the scientific integrity of the study. The study coordinator or principal investigator will follow the IRB's designated procedures for reporting such events or changes and ensure timely communication to the IRB

6. For Non-VCU Sites: For each site or institution listed as "Site Engaged -- Requests to Rely on VCU IRB Review," upload:

Completed Local Context Form for Relying on VCU's IRB

- Site specific informed consent form(s) and HIPAA authorization(s), if applicable

For Foreign Sites: For each Cultural Consultant upload a CV/Biosketch that includes a clear description of cultural expertise:

| | Document<br>Name | Document | Versior | Version Date Upl<br>Wodified By | Uploaded <sub>Type</sub><br>By | Type | Approved |
|---|---|---|---|---|---|---|---|
| | | 02.20.2023.docx | | | | | |
| View | View VS biosketch | Sheppard<br>Biosketch for AN<br>11.14.2022.pdf | 0.01 | 2/20/2023 Asmaa<br>4:00 PM Namoos | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |
| View | Communication<br>log | View Communication Communication log.docx | 0.01 | 2/20/2023 Asmaa<br>3:59 PM Namoos | Asmaa<br>Namoos | Other | Yes |
| View | View PRMC approval 2022-10-10-10-10-10-10-10-10-10-10-10-10-10- | 2022-10-<br>10_MCC-22-<br>19873_PRMC<br>Approval<br>Letter.pdf | 0.01 | 10/10/2022 Asmaa<br>12:30 PM Namoos | Asmaa<br>Namoos | Ancillary Committee<br>Approval | Not<br>Applicable |
| View | View F <b>lye</b> r | Flyer<br>004.08.2022.png | 0.01 | 4/8/2022<br>6:09 PM | Asmaa<br>Namoos | Other | Yes |
| View | View Namoos<br>Resume | Dr. Namoos A.<br>Biosketch<br>06.07.2021.pdf | 0.01 | 4/3/2022<br>3:47 PM | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |

View: SF2 - Personnel

HM20024502 7/8/23, 9:07 AM

ID: HM20024502

### PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

#### Personnel

1. \* List all VCU/VCUHS personnel who are key study personnel.

Key personnel are defined as including: - Conflict of interest investigators, including

- - -the PI
- the Lead Student/Trainee Investigator,
- medically/Psychologically responsible investigator(s)
  - FDA Form 1572 investigators, and
- Other personnel whose roles are essential to the conduct of the research.

Note: Individuals who are not key personnel are not required to be listed here, but PIs still bear the

PIs may elect to use the Study Roster activity button in RAMS-IRB (available after approval) as an alternative way to document study staff involvement and delegation of responsibilities. Personnel changes made to the non-key personnel listed in the separate Study Roster activity do not require an amendment. responsibility to document the delegation of responsibilities in the study records.

| Name Roles | Roles | Roles<br>- Responsibilities - Other<br>Other | Responsibilities Qualifications Qualifications COI - Other Inve | COI<br>Investigator |
|---|---|---|---|---|
| View Tamas<br>Gal | Consultant<br>Co/Sub-Investigator | Data Analysis<br>Data Management<br>Study Design | Experience - Research Education and/or Professional Preparation | yes |
| View Vanessa Consultant<br>Lavene<br>Sheppard Principal Inv<br>Co/Sub-Inve | Vanessa Consultant<br>Lavene<br>Sheppard Principal Investigator<br>Co/Sub-Investigator | Study Design | Experience - Research Experience - Related Skills Education and/or Professional | yes |

| Name | Roles | Roles<br>- Responsibilities Other Qualifications - Other Inve | es Qualifications - Other | ons COI<br>Investigator |
|---|---|---|---|---|
| View Asmaa<br>Namoos | Lead Student/Trainee<br>Investigator (leading<br>their own project)<br>Research Assistant<br>Trainee/Student(working<br>on project) | Data Analysis Project Coordination Data Collection - Direct Observation Participant Consent Data Collection - Lab Regulatory Management Data Management Clinical Participant Identification Data Entry Study Design Data Coding Participant Recruitment Intervention Services Clinical Services Data Collection - Interviews/Surveys | Experience - Research Experience - Related Skills Experience - Clinical Education and/or Professional Preparation Student Trainee | yes |
| View Robert Perera | Consultant<br>Co/Sub-Investigator<br>Statistician | Data Analysis<br>Data Management<br>Data Entry<br>Study Design<br>Data Coding<br>Intervention<br>Services | Experience -<br>Research<br>Education<br>and/or<br>Professional<br>Preparation | yes |
| View Jessica<br>LaRose | Co/Sub-Investigator | Data Analysis<br>Study Design | Experience -<br>Research | yes |

| Name Roles | Roles<br>- Responsibilities Other Qualifications Other Inve | s Qualifications - Other | ns COI<br>Investigator |
|---|---|---|---|
| | Intervention<br>Services | Education<br>and/or<br>Professional<br>Preparation | |
| View Sun Jung Consultant<br>Kim<br>Co/Sub-Investigator | Data Analysis Data Collection - Direct Observation Study Design Data Collection - Interviews/Surveys | Experience - Research Education and/or Professional | yes |

2. Identify all independent investigators and key personnel at non-VCU sites who will be engaged in this study AND who DO NOT have IRB approval for this study from their own institution.

Investigator Other Name Roles -

There are no items to display

- with the research are adequately informed about the protocol and their research related duties and functions: training these individuals will complete and the process that will be used to ensure that all persons assisting 3. If independent investigators or community engaged investigators are listed above, describe the human subjects
- 4. \* Upload a CV or Biosketch for the PI, Medically/Psychologically Responsible Investigators and the lead Student/Trainee Investigators. Do not upload CVs or Biosketches for other individuals.

| Document<br>Name | Document | Versior | Date<br>Modified | Version Modified By | <sup>1</sup> Type | Approved |
|---|---|---|---|---|---|---|
| View Consent form focus group | Namoos- Consent 0.03<br>from of focus<br>group<br>05.12.2023.pdf | t 0.03 | 7/8/2023 Asmaa<br>1:09 AM Namoos | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | n Yes |
| View Consent form - Namoos- Consent 0.04 Intervention from of Intervention group 05.12.2023 copy.pdf | Namoos- Consent<br>from of<br>Intervention group<br>05.12.2023<br>copy.pdf | t 0.04 | 7/8/2023 Asmaa<br>1:09 AM Namoos | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | n Yes |
| View Fund Plan | Asmaa -Budget<br>04.13.2023.xlsx | 0.03 | 5/12/2023 Asmaa<br>11:52 AM Namoos | Asmaa<br>Namoos | Funding Proposal | Not<br>Applicable |

| - | ı | I | | ı | ı | | | | ı | I | ı |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Approved | Yes | Yes | Yes | Yes | Yes | Yes | Yes | ation No | Not<br>Applicable | Yes | Not<br>Applicable |
| Туре | Other | Other | Research Measure | Other | Other | Other | Research Measure | Consent/Assent/Information No<br>Sheet | CV/Biosketch | Other | Ancillary Committee<br>Approval |
| Uploaded <sub>Type</sub><br>By | Asmaa<br>Namoos | Asmaa<br>Namoos | Asmaa<br>Namoos | Asmaa<br>Namoos | Asmaa<br>Namoos | Asmaa<br>Namoos | Asmaa<br>Namoos | Asmaa<br>Namoos | Asmaa<br>Namoos | Asmaa<br>Namoos | Asmaa<br>Namoos |
| Version Date Up | 5/12/2023<br>10:52 AM | 5/12/2023<br>10:43 AM | 5/12/2023<br>10:40 AM | 5/12/2023<br>10:39 AM | 5/12/2023<br>10:24 AM | 5/12/2023<br>6:45 AM | 5/12/2023<br>6:35 AM | 2/20/2023<br>4:32 PM | 2/20/2023<br>4:00 PM | 2/20/2023<br>3:59 PM | 10/10/2022 Asmaa<br>12:30 PM Namoo |
| Version | 0.02 | 0.02 | 0.02 | 0.01 | 0.02 | 0.01 | 0.01 | 0.01 | 0.01 | 0.01 | 0.01 |
| Document | Asmaa Education 0.02 session guide, intervention group-04.07.2023.docx | Namoos, timeline<br>for PROMIS<br>women<br>Projectdocx | Asmaa<br>Conceptual Model<br>05.12.2023.docx | Asmaa Flyer<br>Version<br>05.12.2023.docx | Namoos -Focus<br>Group Script<br>Guide.docx | Namoos-<br>Participants -RA<br>communication<br>script .docx | Survey- Promise<br>women project<br>05.12.2023.docx | Consent from -<br>Focus group<br>02.20.2023.docx | Sheppard<br>Biosketch for AN<br>11.14.2022.pdf | Communication<br>log.docx | 2022-10-<br>10_MCC-22-<br>19873_PRMC<br>Approval |
| Document<br>Name | Education<br>session | View Timeline Plan | Conceptual<br>model | View Flayer 2 | Namoos-Focus<br>group script<br>guide | Participants -RA communication script | Study Survey(<br>Pre-post and<br>satisfactory<br>scales) | consent form-<br>focus group | View VS biosketch | Communication<br>log | PRMC approval |
| | View | View | View | View | View | View | View | View | View | View | View |

| Document<br>Name | Document | Version | Date<br>Modified | Version Date Uploaded Type Modified By | <sup>1</sup> Type | Approved |
|---|---|---|---|---|---|---|
| View Flyer | Flyer<br>004.08.2022.png | 0.01 | 4/8/2022 <i>H</i> 6:09 PM | Asmaa<br>Vamoos | Other | Yes |
| View Namoos<br>Resume | Dr. Namoos A. 0.01<br>Biosketch | 0.01 | 4/3/2022<br>3:47 PM | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |

ID: HM20024502

View: SF2 - Conflict of Interest

### HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN

### Conflict of Interest

The PI should ask the questions on this page of all research personnel who are engaged in the research, including subrecipient investigators and personnel.

1.  $^{\star}$  To the best of your knowledge, do you (as PI) or any other engaged individual have a financial interest related to this study?

consultant, or advisory board member, or officer/director with a related entity; and equity or business Financial interest include utilizing your licensed intellectual property in the study; serving as a paid ownership in a company that is related to this project







 $2.~^{*}$  To the best of your knowledge, do you (as PI) or any other engaged individual have a non-financial interest related to this study?

Non-financial Interests could include such things as:

- utilizing your unlicensed intellectual property in the study,
- serving as an unpaid advisory board member or officer/director with a related entity, and
- equity or business ownership in a company that has yet to make a profit and is related to this project
  - conflict of time/effort,
- personal and professional relationships/affiliations,
- intellectual passions or personal beliefs
- · other factors that could create bias in the study



3. Describe any institutional conflict of interest that you or any member of the research team are aware of that pertains to this research:

An institutional conflict of interest is a situation in which financial interests of the University or University leadership may affect research activities at VCU.

ID: HM20024502

View: SF2 - Other VCU Requirementsv2

### PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

### Other VCU Requirements

This page asks questions on behalf of other ancillary offices, committees and departments at VCU regarding nstitutional requirements that could apply to this research. In some cases, these requirements could also impact the consent process or other aspects of the IRB's review.

Based upon answers provided earlier in this form, certain ancillary sections below may not have questions displayed if those requirements are not applicable to this study.

- 1. Cost Coverage Analysis
- Research Compliance Program at https://research.vcu.edu/human-research/clinical-research/vcu-clinical-research-Information on coverage analysis requirements and processes can be found through VCU's Clinical coverage-analysis/
- required. Has your study been evaluated by an institutionally designated Coverage Analysis Specialist? 1. \* VCU requires that all clinical research studies be evaluated to determine if a Coverage Analysis is
  - Yes
- oN (
- Not Applicable

2. ClinicalTrials.gov Program & OnCore

For guidance, see https://cctr.vcu.edu/support/consultation/clinical-trials-gov/ or email CCTRCTGOV@vcu.edu

- 1. \* Is this a Clinical Trial?

- 2.  $^{*}$  ThePI acknowledges awareness of the following requirements for posting clinical trial consent forms:
- department or agency must post one IRB-approved consent form that was used to enroll subjects on a publicly available Federal website [45 CFR 46.116(h)]. - Each clinical trial under the 2018 Common Rule that is conducted or supported by a Federal
- When engaged in multi-site research, the VCU PI is responsible for confirming with the lead site who is responsible for posting the informed consent form.
  - When VCU is the lead site, the VCU PI is responsible for posting the informed consent form (unless

the federal department or agency will post it).

Yes No

3. Community Engagement

For more information, see https://community.vcu.edu/

1. \* Is this a community engaged research study? (See help text for definitions)

2. \* Provide details about each community co-researcher. If there are more than 5 community partners/coresearchers, add the 5 most significant partners/co-researchers.

| Organization | Zip Code /<br>Country | Role |
|---|---|---|
| Islamic center of<br>Richmond | 23060 | Provides access to study subjects or project sites only. Partner/Coresearcher is not involved with study design, subject recruitment, data collection, or data analysis |

For guidance, see https://rar.vcu.edu/records/family-educational-rights-and-privacy-act/ 4. Family Educational Rights and Privacy Act (FERPA) Requirements

1. \* Does this study involve obtaining information from VCU students' educational records (see help text)?

5. Research Data Privacy Requirements

Contact the VCU Research Data Privacy Office with questions: https://research.vcu.edu/integrity-andcompliance/compliance/research-data-privacy/ 1. \* Does this study involve the VCU site (regardless of the IRB of record), or any sites under the VCU IRB''s oversight, obtaining data in, or from, a foreign country?



#### 6. Information Security

For guidance, see https://ts.vcu.edu/askit/essential-computing/information-security/

1. \* Using the VCU Data Classification Tool, please determine the appropriate data classification category for the data that will be collected or used in this research.

Note: if the data falls into Category 1, a data security management plan is required by University Information Security Office. See help text for information on accessing the VCU Data Classification Tool, and for information on creating a data security management plan at https://dms.vcu.edu. Category 1: all data that require breach notifications in the event of improper release, including Category 2: all proprietary data that if improperly released has the potential to cause harm to the personally identifiable information covered by HIPAA and Commonwealth of Virginia regulations

institution, its mission or its reputation that do not require breach notifications.

2. \* I confirm use of the VCU Data Classification Tool at https://go.vcu.edu/dataclassification in determining the data classification category selected in Question 1:

Yes

2

3. \* The PI is aware that if the study's data is classified as Category 1, a Data Management Plan must be https://ts.vcu.edu/askit/essential-computing/information-security/data-management-system/ submitted to and approved by VCU Information Security prior to IRB approval. See

are maintained external to VCU or hosted by another institution and are NOT currently listed in the DMS system as an approved service for the storage, processing, or transmission of VCU data, I am required study's Data Management Plan. If this study uses any technology platforms, apps, services, etc. that 4. \* I confirm that any use of external technology has been submitted to Information Security in the to have VCU Information Security conduct a security review of that technology. I may contact infosec@vcu.edu with questions.

I also confirm that if the study involves use of external technology and VCUHS HIPAA data, I must also seek security review from the VCUHS Data Governance group (contact Mary Harmon at mary.harmon@vcuhealth.org)

N/A - not using external technology

7. Massey Cancer Center Protocol Review and Monitoring Committee (PRMC) For guidance, see https://www.masseycancercenter.org/research/~/link.aspx? id=ee49e95faa8b44d09b6e89d8e3b48b578\_z=z

- 1. \* Does this study involve any of the following?
- Research involving patients with cancer, their families or their health care providers
  - Research involving cancer screening, diagnosis or prevention
- Secondary data collected from cancer patients or their medical records
- Cancer-related surveys (e.g., attitudes about risk, prevention and treatment) of the general population



If Yes, upload documentation of PRMC approval or review.

- 8. VCU ONETRAC Protocol Review Oversight Committees (PROCs) For guidance, see https://onetrac.vcu.edu/
- 1. \* Does this study involve research with any of the following?
- VCU Health System patients
- VCU Health System facilities
- VCU Health System data



Yes

9. VCU Health Department of Patient Centered Services

- 1. \* Does your study involve a satisfaction survey administered to VCUHS patients (\*See Help Text):
- ŝ

Not Applicable

10. VCU Faculty-Held IND or IDE

For guidance, see https://research.vcu.edu/human-research/regulatory-affairs/.

Questions related to if you need an IND or IDE for your study should be emailed to: indide@vcu.edu. Please submit a

copy of your FDA submitting to the FDA to https://redcap.vcu.edu/surveys/?s=NR7K7LR4JW.

### 11. VCU Health System locations

| Will research ommunity Me | <b>ხ</b> | emorial Hospital, Tappahannock Hospital, VCU Medical Center and Massey Cancer | |
|---|---|---|---|
| * O C | Will research activities occu | al Hospi | Centerl? |



12. VCUHS Department of Pathology

ŝ

Learn more about requesting and establishing an account with Pathology here: See https://pathology.vcu.edu/research-services/

- 1. \* I have contacted VCUHS Department of Pathology to determine feasibility if my study involves the following:
  - Storage of Microbiology isolates
- New instrumentation provided by clinical trial/study sponsor, or
- Non-routine specimen processing (examples include but aren't limited to the following: addition of reagents to samples/aliquots, buffy coat processing, DNA sample processing)

| (O | |
|-----|---|
| Yes | |
| | ر |



N/A - my study does not involve any of the listed processes.

- 2. \* If my study involves specimen retrieval from the Pathology laboratory, I have established a process with Pathology to deidentify and retrieve specimens.
- Xes C
- §

N/A - my study won't involve specimen retrieval from Pathology

13. VCU Institutional Biosafety Committee (IBC)

To contact the Biosafety Office see their website at: https://research.vcu.edu/integrity-andcompliance/compliance/regulatory-committees/

that have NOT been FDA approved? These may include, but are not limited to, any of the following. If 1. \* Does this project involve any of the following hazardous biological agents ("biohazardous agents") you are unsure, please contact the Biosafety Office:  - Any functional recombinant viruses (especially viruses that may integrate into the patients' genome).

- Expression or administration of biological toxins.
- Live pathogenic or potentially pathogenic organisms of plants or animals (bacteria, fungi, wildtype viruses, parasites, etc.), that are, or potentially may be, in experimental products.
- Introduction or expression of rDNA or synthetic nucleic acids
- Use of a product (e.g., monoclonal antibodies, recombinant cytokines) produced from virally infected mammalian cells.
- Use of a product (purified growth factors, cytokines) produced from mammals or their cells.



14. VCU Radiation Safety Committee (RSC)

To contact the Radiation Safety Section see their website at: https://research.vcu.edu/integrity-andcompliance/compliance/regulatory-committees/

- 1. \* Does this study involve radiation exposure and/or scans involving radiation (e.g.: PET, MRA, CT, DXA, nuclear medicine, etc.)?
- ) Yes
- 15. VCU Scientific Review Committee (SRC)

For guidance, see https://cctr.vcu.edu/support/consultation/scientific-review-committee/

- 1. \* Has this human subjects protocol (not the grant application) already been reviewed by the funder of a sponsored project (e.g. a federal, state or non-profit funding sponsor)?

16. Upload any documents requested in the questions above:

| CC991CBE9AD565000?packetIds=defaultPrintPacket |
|------------------------------------------------|
| 1EC |
| 4A9571 |
| B0E834 |
| / |
| Protoco |
| ject/ |
| ıtPro |
| n/prir |
| rtforr |
| /sma |
| ortal |
| app/p |
| ı/irb/ |
| u.edı |
| ch.vcu |
| researd |
| /irb.r |
| https:/ |

| | Document<br>Name | Document | Versior | Version Date Upl<br>Modified By | Uploaded <sub>Type</sub><br>By | Туре | Approved |
|---|---|---|---|---|---|---|---|
| | | 02.20.2023.docx | | | | | |
| View | View VS biosketch | Sheppard<br>Biosketch for AN<br>11.14.2022.pdf | 0.01 | 2/20/2023<br>4:00 PM | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |
| View | View Communication Communication log log.docx | Communication log.docx | 0.01 | 2/20/2023 Asmaa<br>3:59 PM Namoos | Asmaa<br>Namoos | Other | Yes |
| View | View PRMC approval 2022-10-10-10-10-10-10-10-10-10-10-10-10-10- | 2022-10-<br>10_MCC-22-<br>19873_PRMC<br>Approval<br>Letter.pdf | 0.01 | 10/10/2022 Asmaa<br>12:30 PM Namoos | Asmaa<br>Namoos | Ancillary Committee<br>Approval | Not<br>Applicable |
| View | View Flyer | Flyer<br>004.08.2022.png | 0.01 | 4/8/2022<br>6:09 PM | Asmaa<br>Namoos | Other | Yes |
| View | View Namoos<br>Resume | Dr. Namoos A.<br>Biosketch<br>06.07.2021.pdf | 0.01 | 4/3/2022<br>3:47 PM | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |

HM20024502 ID: HM20024502

View: SF2 - Institutional Requirements Complete

PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn HM20024502 - Vanessa Lavene Sheppard methods among Muslim Americans WOMEN

# Institutional Requirements Complete

Protocol Progress:

- **INITIAL SETUP**
- **BACKGROUND, RATIONALE & GOALS**
- **RESEARCH PLAN**
- CONSENT PLAN
- RISKS, PRIVACY & CONFIDENTIALITY
- POPULATIONS WITH SPECIAL CONSIDERATIONS
  - INSTITUTIONAL REQUIREMENTS® DOCUMENTS

Click Continue below to go to the next section

View: SF2 - Documents HM20024502

ID: HM20024502

7/8/23, 9:07 AM

### HM20024502 - Vanessa Lavene Sheppard PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN

#### **Documents**

1. Upload any documents that the VCU IRB will need to conduct a review of this submission: A list of potential documents is given in the help text NOTE: The delete function should only be used if an incorrect document is uploaded or added to the system AND that document has not been reviewed and approved by the IRB. Do NOT delete documents that the IRB previously reviewed and approved.

the same document) should be added to the IRB submission by using the Update button. To provide updated Once you have uploaded a document to RAMS-IRB, any changes to that document (i.e. different versions of documents, follow these steps:

- Click the Update button located to the left of the document to be updated.
- In the Add Document window, click the Choose File or Browse button, select the file you are adding, and click on the Open button.
- Click OK to close the Add Document window, and the system will upload the revised document. RAMS-IRB will automatically provide a version number for the document.

To access previous versions of a document in RAMS-IRB you must use the History link associated with the

- Click the View or Update button located to the left of the document you wish to access.
- In the Add/View Document window, click the "History" hyperlink located to the right of the file name.
- A separate window will open that shows all versions of the document that have been added to RAMS-IRB. Click on any file name to download and view the document.

| Document<br>Name | Document | Version | )ate<br>Nodified | Version Modified By | | Approved |
|---|---|---|---|---|---|---|
| View Consent form focus group | Namoos- Consent 0.03<br>from of focus<br>group<br>05.12.2023.pdf | | 7/8/2023<br>1:09 AM | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | , es |
| View Consent form Intervention program | View Consent form - Namoos- Consent 0.04 Intervention from of Intervention group 05.12.2023 copy.pdf | | 7/8/2023 Asmaa<br>1:09 AM Namoos | Asmaa<br>Namoos | Consent/Assent/Information Yes<br>Sheet | , es |
| View Fund Plan | Asmaa -Budget<br>04.13.2023.xlsx | 0.03 | 5/12/2023 Asmaa<br>11:52 AM Namoos | Asmaa<br>Namoos | Funding Proposal A | Not<br>Applicable |

| | Document<br>Name | Document | Version | Date<br>Modified | Version Date Uploaded Type Modified By | <sup>1</sup> Type | Approved |
|---|---|---|---|---|---|---|---|
| View | /iew Flyer | Flyer<br>004.08.2022.png | 0.01 | 4/8/2022<br>6:09 PM | Asmaa<br>Namoos | Other | Yes |
| View | Namoos<br>Resume | Dr. Namoos A.<br>Biosketch<br>06.07.2021.pdf | 0.01 | 4/3/2022<br>3:47 PM | Asmaa<br>Namoos | CV/Biosketch | Not<br>Applicable |

ID: HM20024502

View: SF2 - Documents Complete

PROMIS WOMAN Education Program: ImProving ceRvical cancer preventiOn methods among Muslim Americans WOMEN HM20024502 - Vanessa Lavene Sheppard

### Documents Complete

Protocol Progress:

**● INITIAL SETUP** 

**BACKGROUND, RATIONALE & GOALS** 

RESEARCH PLAN

CONSENT PLAN

RISKS, PRIVACY & CONFIDENTIALITY

POPULATIONS WITH SPECIAL CONSIDERATIONS

INSTITUTIONAL REQUIREMENTS

DOCUMENTS

End of Application

Click Continue below to exit and submit this project

View: SF\_IRB\_ConsentPlan\_Groups

7/8/23, 9:07 AM

HM20024502

### Consent Groups

| :dno | |
|--------------------------------------|-------------------|
| gro | |
| ent | |
| ass | |
| 'n. | |
| nse | |
| ၁၁ | |
| ŧ | |
| for | |
| name for this consent / assent group | Ę |
| ē | 횬 |
| pti | onsen |
| a descripti | ŝ |
| de | dno |
| era | cus gr |
| Ent | ocus group consen |
| * | т |

| * S | <u>elec</u> | * Select all that apply to this consent / assent group: |
|---|---|---|
| | | Name |
| | | Signed Consent by Participant |
| | | Signed Parent/Guardian Permission or Legally Authorized Representative Consent |
| | | Signed Assent by Child or Decisionally Impaired Adult |
| | | Verbal/Other Indication of Assent by Child or Decisionally Impaired Adult |
| | | Short Form Consent (limited applicability) |
| | | None of the Above (select waiver below) |
| χ.<br>Υ. | ĕ ☐ | * Select all electronic signature platforms that apply to this consent / assent group: Not using electronic signature platforms |
| | | DocuSign Part 11 (FDA regulated studies) |
| | > | DocuSian (standard platform for non-FDA regulated studies) |

iMedConsent (Veterans Affairs studies)

REDCap e-Consent

Other electronic signature platform

5. \* Select any waivers that apply to this consent / assent group:

| > | No Waivers Requested |
|---|---|
| | Waiver of All Consent or Some Elements in Consent Form |
| | Waiver of Parental Permission or Legally Authorized Representative Consent |
| | Waiver of All Assent by Child or Decisionally Impaired Adult |
| | Waiver of Signature on Consent/Permission Forms (waiver of documentation of consent) |
| | Exception from Informed Consent (for emergency research only) |
| s, * Selec | 6. * Select all study team role(s) that will obtain consent / assent from this group: |
| > | Principal Investigator |
| > | Co/Sub-Investigator |
| | Medical or Psychological Responsible Investigator |
| > | Lead Student/Trainee Investigator (leading their own project) |
| > | Research Coordinator |
| | Research Nurse |
| | Consultant |

| Research Assistant |
|-------------------------------------|
| Pharmacist |
| Statistician |
| Regulatory Coordinator |
| Trainee/Student(working on project) |
| Other |
| N/A: Requesting Waiver of Consent |

- 7. \* Describe the consent procedures used for this group. Address each point below:
- When and where consent will occur
- What will be covered during the consent discussion
- How the consent discussion will occur (e.g. in-person, phone, video conference)
  - How you will reconfirm consent on an ongoing basis, if applicable

participants will be provided with a background about cervical cancer among Muslim women. Depending on their -The consenting process for the study will commence after receiving IRB approval, expected in May 2023, at the enrollment, either in the focus group or the education session, the details of the respective components will be Islamic Center in a private room provided by the Community Advisory Board. During the consent discussion,

-The consent discussion will take place in-person, allowing for face-to-face interaction. The research assistant (RA) will provide the participant with the necessary materials and information to make an informed decision about participation. The discussion will cover the potential risks, benefits, and compensation associated with the study.

-Participants will be given the opportunity to consider their participation and make an informed decision. They will be offered the option to provide consent electronically using either DocuSign. The electronic consent form will be accessible via a provided link, ensuring convenience and ease of use for the participants.

- Ongoing reconfirmation of consent is not applicable in this study.
- $8 \cdot *$  Select the processes for minimizing any potential perception of undue influence to participate, particularly when there is a pre-existing relationship between the participant and the researcher (e.g. treatment

provider/patient; instructor/student; supervisor/employee, etc.):

### 9. \* Describe the other ways the study team will minimize any potential perception of undue influence to participate:

our team is supported by the Mosque and our names and pictures will be on the Ads board to make sure we are Our team will offer enough privacy to let the Muslim women think and join to our study. trusted by the community.

## 10. \* How much time will participants be given to make a decision:

Two weeks after the first conversation about the study, we will drop the participant from out list if we have not heard back from her 11. If applicable, describe the procedures for consenting children upon entering adulthood or participants who are no longer decisionally impaired:
# Consent Groups

| this consent / assent group: | |
|-------------------------------------|---------------------------------|
| 1. * Enter a descriptive name for t | Intervention group consent form |

| assent group: |
|---------------|
| _ |
| consent |
| js |
| Ξ |
| $\overline{}$ |
| ¥ |
| ıt apply |
| at |
| 읖 |
| = |
| a |
| ದ್ದ |
| 픚 |
| Select |
| * |
| ď |

| | Name |
|---|---|
| > | Signed Consent by Participant |
| | Signed Parent/Guardian Permission or Legally Authorized Representative Consent |
| | Signed Assent by Child or Decisionally Impaired Adult |
| | Verbal/Other Indication of Assent by Child or Decisionally Impaired Adult |
| | Short Form Consent (limited applicability) |
| | None of the Above (select waiver below) |
| 3. * Selec | * Select all electronic signature platforms that apply to this consent / assent group: |
| | Not using electronic signature platforms |
| | DocuSign Part 11 (FDA regulated studies) |
| > | DocuSign (standard platform for non-FDA regulated studies) |
| | REDCap e-Consent |

iMedConsent (Veterans Affairs studies)

Other electronic signature platform

4. If Other is selected, explain:

7/8/23, 9:07 AM

5. \* Select any waivers that apply to this consent / assent group:

| > | No Waivers Requested |
|---|---|
| | Waiver of All Consent or Some Elements in Consent Form |
| | Waiver of Parental Permission or Legally Authorized Representative Consent |
| | Waiver of All Assent by Child or Decisionally Impaired Adult |
| | Waiver of Signature on Consent/Permission Forms (waiver of documentation of consent) |
| | Exception from Informed Consent (for emergency research only) |
| 6, * Selec | 6. * Select all study team role(s) that will obtain consent / assent from this group: |
| > | Principal Investigator |
| | Co/Sub-Investigator |
| | Medical or Psychological Responsible Investigator |
| > | Lead Student/Trainee Investigator (leading their own project) |
| > | Research Coordinator |
| | Research Nurse |
| | Consultant |

| > | Research Assistant |
|---|-------------------------------------|
| | Pharmacist |
| | Statistician |
| | Regulatory Coordinator |
| > | Trainee/Student(working on project) |
| | Other |
| | N/A: Requesting Waiver of Consent |

# 7. \* Describe the consent procedures used for this group. Address each point below:

- When and where consent will occur
- What will be covered during the consent discussion
- How the consent discussion will occur (e.g. in-person, phone, video conference)
  - How you will reconfirm consent on an ongoing basis, if applicable

When and Where Consent Will Occur:

Consent for the intervention group will be obtained at the Islamic Center during the scheduled education sessions. Participants will have the opportunity to provide consent before engaging in the educational program.

What Will Be Covered During the Consent Discussion:

confidentiality and the voluntary nature of their involvement. They will have the opportunity to ask questions and seek participation will be clearly explained, along with any potential discomfort or adverse effects that may arise from the educational sessions. Additionally, participants will be informed about their rights as research participants, including During the consent discussion, participants will be provided with a detailed explanation of the educational program, including the topics covered, session duration, and expected outcomes. The risks and benefits associated with clarifications before providing consent.

How the Consent Discussion Will Occur:

participants. A designated research team member, such as the research assistant (RA), will conduct the discussion in a provide explanations and guidance as needed to ensure the participant's understanding of the study and their role in it. questions, and discuss any concerns before making an informed decision to participate. The RA will be available to The consent discussion will occur in-person, allowing for direct communication between the research team and the private room at the Islamic Center. The participant will have the opportunity to review the consent form, ask any

withdraw from the study at any time, even after providing initial consent. Participants will also be provided with contact information to reach out to the research team if they have any questions or concerns during or after the educational Since the intervention group will be participating in a one-day educational program, ongoing reconfirmation of consent is not applicable in this case. However, the research team will ensure that participants are aware of their right to How Consent Will Be Reconfirmed on an Ongoing Basis: program.

œ̈

| Selec<br>when the | Select the processes for minimizing any potential perception of undue influence to participate, particularly when there is a pre-existing relationship between the participant and the researcher (e.g. treatment provider/patient; instructor/student; supervisor/employee, etc.): Having a 3rd person (family/friends, another study team member, etc.) present during the consent / assent |
|---|---|
| | discussion |
| | Having an independent advocate (e.g. advocate for decisionally impaired adults, wards) present during the consent / assent discussion |
| | Removing physical symbols of authority like white coats or police badges |
| | Sitting down beside the participant instead of standing over them |
| | If obtaining consent / assent in a clinical setting, letting patients sit instead of lie down (if they are able to) |
| | Moving to a more neutral location like a conference room |
| | Obtaining consent / assent after other services/interactions have been completed (e.g. after school or the clinic visit) |
| > | Having a mandatory wait period for the participant to go home and think before they sign consent<br><i>l</i> assent |
| | Sharing the consent / assent discussion between two people (i.e. a clinician might be the best person to explain study procedures and risks, but then they could step out and let a research assistant finish the consent process) |
| | Other protection(s) not listed here – describe below |
| | N/A: Requesting Waiver of Consent |

9. \* Describe the other ways the study team will minimize any potential perception of undue influence to participate:

First, participants will be provided with comprehensive information about the study, including its purpose, procedures, risks, benefits, and their rights as research participants. This will allow them to make an informed decision based on To minimize any potential perception of undue influence to participate, the study team will employ various strategies. heir own judgment.

Second, the study team will ensure that participation is voluntary, and participants can choose to withdraw from the study at any time without consequences.

Third, the consent process will be conducted in a private and comfortable setting, allowing participants to freely express their concerns and ask questions.

reach out for further clarification or to voice any concerns they may have throughout the study. These measures aim to Finally, the study team will maintain open lines of communication and provide contact information so participants can create a supportive and unbiased environment, promoting autonomy and safeguarding against perceived undue influence.

# 10. \* How much time will participants be given to make a decision:

Participants will be given sufficient time (expecting from a week to two weeks) to make a decision regarding their participation in the study. The exact duration may vary depending on the circumstances and complexity of the study. Typically, participants are encouraged to take as much time as they need to review the provided information, ask questions, and consider their decision.

The study team will emphasize that there is no rush to make a decision and that participants are free to take the necessary time to make an informed choice that aligns with their interests and preferences. 11. If applicable, describe the procedures for consenting children upon entering adulthood or participants who are no longer decisionally impaired:

7/8/23, 9:07 AM ID: HM20024502 **HM20024502**  View: SF\_IRB\_StudyLocation\_NonVCUSitesDetails

# Non-VCU Site Details

- 1. \* Name of institution or site:
  - The University of Kentucky
- performing. For example involvement in study design, carrying out research procedures, recruiting subjects, 2. \* Provide a description of the institution's or site's role in the research and what study activities they will be consenting, analyzing data and or specimens (regardless of identifiability), writing manuscripts or publications, solely being a location for VCU investigators to conduct activities, etc.:
  - The University of Kentucky (UK) collaborates with VCU investigators by actively participating in research studies. Their role may observing the recruitment process and contributing to manuscript writing. They are not solely a location for VCU investigators but actively engage in various research activities.
- 3. \* Describe the adequacy of the institution or site to ensure human participant safety, particularly in event of institution, ensures that appropriate measures are in place to protect the safety and well-being of participants in the In the context of research conducted at VCU collaboration with the University of Kentucky (UK),human participant safety will be observed by VCU and overseen by their Institutional Review Board (IRB). VCU, as the responsible event of an unanticipated emergency. unanticipated emergency:

The VCU IRB provides oversight and guidance to ensure that all necessary precautions are taken to safeguard the participants throughout the research process.

| :wc |
|----------|
| ill folk |
| site w |
| tion or |
| institu |
| UDV- |
| ne Nor |
| path th |
| eview |
| BB r |
| lect the |
| * Se |

| Exempt study submission |
|---|
| Site Engaged Has FWA and Will Obtain Own IRB Review |
| Site Engaged Requests to Rely on VCU IRB Review |
| Site Not Engaged IRB Review Not Required |
| Site Engaged Does not regularly conduct human subject research AND is not required to have a FWA as a recipient of PHS funding. |

113/155

- 5. If the institution or site is engaged and will either 1) obtain their own IRB review OR 2) rely on VCU IRB review, provide the FWA# of the site:
- 6. If this is a foreign site or location, select which individuals and/or groups will be serving as the cultural consultant for the site to ensure that the research will be conducted according to local customs and procedures:
- This is not a foreign site/location
- Foreign IRB or ethics committee (required for foreign sites engaged in expedited and full board research)
- Foreign site principal investigator
- Foreign site community advisory board
- Foreign site community elders or similar governing body
- Other cultural consultant (select if none of the above options apply; more information will be required about this individual)

ID: HM20024502

View: Personnel

#### Personnel

| | ( |
|---|---|
| Φ | • |
| | - |
| ᇤ | - |
| ಹ | |
| Ź | |
| < | ŀ |
| _ | |
| • | |

Tamas Gal

2. \* Is this individual a 'COI Investigator'?

Conflict of Interest (COI) Investigator - any individual who has a level of independence and responsibility comparable to that of the PI for the design, conduct, or reporting of research.

Anyone designated as a COI Investigator must have a current Financial Interest Report (FIR) in the Activity and Interest Reporting System (AIRS) (https://airs.research.vcu.edu).

| | | | | ısible Investigator | or (leading their own project) | | | |
|---|---|---|---|---|---|---|---|---|
| Yes | es: | Principal Investigator | Co/Sub-Investigator | Medical or Psychological Responsible Investigator | Lead Student/Trainee Investigator (leading their own project) | Research Coordinator | Research Nurse | Consultant |
| | 3. * Roles: | | > | | | | | > |

| | Research Assistant |
|------------|--------------------------------------|
| | Pharmacist |
| | Statistician |
| | Regulatory Coordinator |
| | Trainee/Student(working on project) |
| | Other |
| 4. * Study | 4. * Study related responsibilities: |
| > | Study Design |
| | Data Collection - Lab |
| | Data Collection - Clinical |
| | Data Collection - Interviews/Surveys |
| | Data Collection - Direct Observation |
| | Clinical Services |
| | Intervention Services |
| | Data Entry |

| Data Coding |
|---|
| Data Management |
| Data Analysis |
| Project Coordination |
| Participant Identification |
| Participant Recruitment |
| Participant Consent |
| Regulatory Management |
| Other |
| <ol> <li>The PI certifies that if this individual will conduct any clinical activities as part of this study, the individual is appropriately credentialed and privileged to practice within the institution where the research will be conducted: Individual has no clinical responsibilities</li> </ol> |
| 6. * Qualifications to carry out study related responsibilities: (you may select multiple answers) |
| Education and/or Professional Preparation |
| Experience - Research |
| Experience - Clinical |
| Experience - Related Skills |

| | | | Emergency Phone: | https://irb.research.vcu.edu/irb/app/portal/smartform/printProject/_Protocol/7B0E8344A95711ECC991CBE9AD565000?packetIds=defaultPrintPacket |
|---|---|---|---|---|
| Trainee | Student | Other | 7. Additional or Emerge | https://irb.research.vcu.edu/irb/app |

ID: HM20024502

7/8/23, 9:07 AM

View: Personnel

#### Personnel

1. \* Name: Vanessa Lavene Sheppard

2. \* Is this individual a 'COI Investigator'?

Conflict of Interest (COI) Investigator - any individual who has a level of independence and responsibility comparable to that of the PI for the design, conduct, or reporting of research.

Anyone designated as a COI Investigator must have a current Financial Interest Report (FIR) in the Activity and Interest Bonorting System (AIBS) (https://pire.googe/housedd)

| Yes No No Co/Sub-Investigator Medical or Psychological Responsible Investigator Lead Student/Trainee Investigator (leading their own projector) Research Nurse Consultant |
|---|
|---|

Research Assistant

7/8/23, 9:07 AM

Pharmacist

Statistician

| Regulatory Coordinator | Trainee/Student(working on project) |
|------------------------|-------------------------------------|

| Other |
|-------|

| (J) |
|---------------|
| (D) |
| .≖ |
| ± |
| ≔ |
| -= |
| _ |
| ທ |
| ≂ |
| Q |
| ğ |
| ī |
| 31 |
| Ψ |
| _ |
| $\overline{}$ |
| ਦ |
| O |
| _ |
| σ |
| 7 |
| ø |
| _ |
| _ |
| 2 |
| 7 |
| 三 |
| 'n |
| υ, |
| * |
| <del>-</del> |
| 7 |

| <b>&gt;</b> |
|-------------|

| Study Design |
|--------------|
| > |

Data Collection - Lab

| חששום סחשבווח |
|---------------|

| Data Collection - Interviews/Surveys | Data Collection - Direct Observation |
|--------------------------------------|--------------------------------------|

| Clinical Services |
|-------------------|
| 1 |

| Intervention Services |
|-----------------------|

| <br>Data Entry |
|----------------|

| ét |
|--------------------------------------------------------------------|
| × |
| ਠ |
| Œ |
| 뒫 |
| Ħ |
| ·≡ |
| <u>ā</u> |
| 표 |
| П |
| ault |
| 75 |
| ŏ |
| ĭĬ |
| S |
| О |
| etId |
| 중 |
| ĕ |
| õ |
| ~ |
| 00 |
| 565000? |
| 5650 |
| ιĊ |
| 92 |
| 9AD |
| ⋖ |
| <u>ത്</u> |
| Щ̈ |
| CB |
| 1CB |
| Ť |
| Ō |
| 6 |
| ECC99 |
| Ö |
| ш |
| ш |
| = |
| 4A957 |
| Ωi |
| 95 |
| ⋖ |
| 4 |
| 4 |
| ന |
| 8 |
| 0E83 |
| 0 |
| //B |
| _ |
| $\overline{}$ |
| 0 |
| 0 |
| 0 |
| rotocol |
| Protoco |
| Protoco |
| rotoco |
| Protoco |
| ect/_Protoco |
| Protoco |
| roject/_Protoco |
| ect/_Protoco |
| Project/_Protoco |
| Project/_Protoco |
| Project/_Protoco |
| Project/_Protoco |
| Project/_Protoco |
| orm/printProject/_Protoco |
| Project/_Protoco |
| orm/printProject/_Protoco |
| rtform/printProject/_Protoco |
| rtform/printProject/_Protoco |
| smartform/printProject/_Protoco |
| al/smartform/printProject/_Protoco |
| rtal/smartform/printProject/_Protoco |
| al/smartform/printProject/_Protoco |
| rtal/smartform/printProject/_Protoco |
| rtal/smartform/printProject/_Protoco |
| rtal/smartform/printProject/_Protoco |
| 'app/portal/smartform/printProject/_Protoco |
| 'app/portal/smartform/printProject/_Protoco |
| rtal/smartform/printProject/_Protoco |
| /irb/app/portal/smartform/printProject/_Protoco |
| u/irb/app/portal/smartform/printProject/_Protoco |
| u/irb/app/portal/smartform/printProject/_Protoco |
| .edu/irb/app/portal/smartform/printProject/_Protoco |
| .edu/irb/app/portal/smartform/printProject/_Protoco |
| cu.edu/irb/app/portal/smartform/printProject/_Protoco |
| search.vcu.edu/irb/app/portal/smartform/printProject/_Protoco |
| cu.edu/irb/app/portal/smartform/printProject/_Protoco |
| search.vcu.edu/irb/app/portal/smartform/printProject/_Protoco |
| rb.research.vcu.edu/irb/app/portal/smartform/printProject/_Protoco |
| search.vcu.edu/irb/app/portal/smartform/printProject/_Protoco |
| rb.research.vcu.edu/irb/app/portal/smartform/printProject/_Protoco |

| HM20024502 |
|-----------------|
| 'AM |
| 7/8/23, 9:07 AM |

| Trainee | Student | Other |
|---------|---------|-------|

7. Additional or Emergency Phone:

ID: HM20024502

View: Personnel

#### Personnel

| | 0 |
|-----|-------|
| | 7 |
| me: | ממ |
| Ē | Asmaa |
| k | ⋖ |
| Ċ | |

2. \* Is this individual a 'COI Investigator'?

Conflict of Interest (COI) Investigator - any individual who has a level of independence and responsibility comparable to that of the PI for the design, conduct, or reporting of research.

Anyone designated as a COI Investigator must have a current Financial Interest Report (FIR) in the Activity and Interest Reporting System (AIRS) (https://airs.research.vcu.edu).

| | Yes |
|-------------|---------------------------------------------------------------|
| 0 | ON ( |
| 3, * Roles: | |
| | Principal Investigator |
| | Co/Sub-Investigator |
| | Medical or Psychological Responsible Investigator |
| > | Lead Student/Trainee Investigator (leading their own project) |
| | Research Coordinator |
| | Research Nurse |
| | Consultant |

| > | Research Assistant |
|----------|--------------------------------------|
| | Pharmacist |
| | Statistician |
| | Regulatory Coordinator |
| > | Trainee/Student(working on project) |
| | Other |
| 4, * Stu | 4. * Study related responsibilities: |
| > | Study Design |
| > | Data Collection - Lab |
| > | Data Collection - Clinical |
| > | Data Collection - Interviews/Surveys |
| > | Data Collection - Direct Observation |
| > | Clinical Services |
| > | Intervention Services |
| > | Data Entry |

| | Data Coding |
|---|---|
| > | Data Management |
| > | Data Analysis |
| > | Project Coordination |
| > | Participant Identification |
| > | Participant Recruitment |
| > | Participant Consent |
| > | Regulatory Management |
| | Other |
| * The<br>appro<br>condi<br>Indivic | 5. * The PI certifies that if this individual will conduct any clinical activities as part of this study, the individual is appropriately credentialed and privileged to practice within the institution where the research will be conducted: Individual has no clinical responsibilities |
| * Qua | 6. * Qualifications to carry out study related responsibilities: (you may select multiple answers) |
| > | Education and/or Professional Preparation |
| > | Experience - Research |
| > | Experience - Clinical |
| > | Experience - Related Skills |

| | Trainee |
|---|---------|
| > | |
| > | Student |
| | Other |

7. Additional or Emergency Phone:

ID: HM20024502

7/8/23, 9:07 AM

View: Personnel

#### Personnel

| | _ |
|-------|---|
| | ā |
| | ā |
| <br>• | Δ |
| യ | |
| Ē | t |
| Ξ | ā |
| ਕ | ~ |
| ž | - |
| _ | C |
| k | Ω |
| _ | |
| - | |

nopert Perera

2. \* Is this individual a 'COI Investigator'?

Conflict of Interest (COI) Investigator - any individual who has a level of independence and responsibility comparable to that of the PI for the design, conduct, or reporting of research.

Anyone designated as a COI Investigator must have a current Financial Interest Report (FIR) in the Activity and Interest Reporting System (AIRS) (https://airs.research.vcu.edu).

| | Yes |
|-------------|---------------------------------------------------------------|
| | ON O |
| 3. * Roles: | les: |
| | Principal Investigator |
| > | Co/Sub-Investigator |
| | Medical or Psychological Responsible Investigator |
| | Lead Student/Trainee Investigator (leading their own project) |
| | Research Coordinator |
| | Research Nurse |
| > | Consultant |

| | Research Assistant |
|--------|--------------------------------------|
| | Pharmacist |
| > | Statistician |
| | Regulatory Coordinator |
| | Trainee/Student(working on project) |
| | Other |
| * Stuc | 4. * Study related responsibilities: |
| > | Study Design |
| | Data Collection - Lab |
| | Data Collection - Clinical |
| | Data Collection - Interviews/Surveys |
| | Data Collection - Direct Observation |
| | Clinical Services |
| > | Intervention Services |
| > | Data Entry |

| | Data Coding |
|---|---|
| > | |
| > | Data Management |
| > | Data Analysis |
| | Project Coordination |
| | Participant Identification |
| | Participant Recruitment |
| | Participant Consent |
| | Regulatory Management |
| | Other |
| * The<br>appro<br>condt<br>Indivic | 5. * The PI certifies that if this individual will conduct any clinical activities as part of this study, the individual is appropriately credentialed and privileged to practice within the institution where the research will be conducted: Individual has no clinical responsibilities |
| . * Qua | 6. * Qualifications to carry out study related responsibilities: (you may select multiple answers) |
| > | Education and/or Professional Preparation |
| > | Experience - Research |
| | Experience - Clinical |
| | Experience - Related Skills |

| COLFICOCOLFIC | 1/45 | 1001 |
|---------------|------|------|

7. Additional or Emergency Phone:

ID: HM20024502

View: Personnel

#### Personnel

| | c |
|---|-----|
| | ď |
| | _ |
| Ĕ | 000 |
| Z | 90 |
| _ | |

Jessica LaRose

2. \* Is this individual a 'COI Investigator'?

Conflict of Interest (COI) Investigator - any individual who has a level of independence and responsibility comparable to that of the PI for the design, conduct, or reporting of research.

Anyone designated as a COI Investigator must have a current Financial Interest Report (FIR) in the Activity and Interest Reporting System (AIRS) (https://airs.research.vcu.edu).

| | Yes |
|-------------|---------------------------------------------------------------|
| O | ON ( |
| 3. * Roles: | :S: |
| | Principal Investigator |
| > | Co/Sub-Investigator |
| | Medical or Psychological Responsible Investigator |
| | Lead Student/Trainee Investigator (leading their own project) |
| | Research Coordinator |
| | Research Nurse |
| | Consultant |

| | Research Assistant |
|-----------|--------------------------------------|
| | Pharmacist |
| | Statistician |
| | Regulatory Coordinator |
| | Trainee/Student(working on project) |
| | Other |
| 4. * Stud | 4. * Study related responsibilities: |
| > | Study Design |
| | Data Collection - Lab |
| | Data Collection - Clinical |
| | Data Collection - Interviews/Surveys |
| | Data Collection - Direct Observation |
| | Clinical Services |
| > | Intervention Services |
| | Data Entry |

| Data Coding |
|---|
| Data Management |
| Data Analysis |
| Project Coordination |
| Participant Identification |
| Participant Recruitment |
| Participant Consent |
| Regulatory Management |
| Other |
| <ol> <li>The PI certifies that if this individual will conduct any clinical activities as part of this study, the individual is appropriately credentialed and privileged to practice within the institution where the research will be conducted: Individual has no clinical responsibilities</li> </ol> |
| 6. * Qualifications to carry out study related responsibilities: (you may select multiple answers) |
| Education and/or Professional Preparation |
| Experience - Research |
| Experience - Clinical |
| Experience - Related Skills |

| S |
|---------------|
| $\dot{\circ}$ |
| ī |
| ₹ |
| Ñ |
| ñ |
| 2 |
| -> |
| = |
| ㅗ |

ID: HM20024502

View: Personnel

#### Personnel

1. \* Name: Sun Jung Kim

2. \* Is this individual a 'COI Investigator'?

Conflict of Interest (COI) Investigator - any individual who has a level of independence and responsibility comparable to that of the PI for the design, conduct, or reporting of research.

Anyone designated as a COI Investigator must have a current Financial Interest Report (FIR) in the Activity and Interest Reporting System (AIRS) (https://airs.research.vcu.edu).

| | | | | l Responsible Investigator | vestigator (leading their own project) | | | |
|---|---|---|---|---|---|---|---|---|
| Yes<br>No | :S: | Principal Investigator | Co/Sub-Investigator | Medical or Psychological Responsible Investigator | Lead Student/Trainee Investigator (leading their own project) | Research Coordinator | Research Nurse | Consultant |
| | 3, * Roles: | | > | | | | | > |

| | Research Assistant |
|----------|--------------------------------------|
| | Pharmacist |
| | Statistician |
| | Regulatory Coordinator |
| | Trainee/Student(working on project) |
| | Other |
| . * Stuc | 4. * Study related responsibilities: |
| > | Study Design |
| | Data Collection - Lab |
| | Data Collection - Clinical |
| > | Data Collection - Interviews/Surveys |
| > | Data Collection - Direct Observation |
| | Clinical Services |
| | Intervention Services |
| | Data Entry |

| Data Coding |
|---|
| Data Management |
| Data Analysis |
| Project Coordination |
| Participant Identification |
| Participant Recruitment |
| Participant Consent |
| Regulatory Management |
| Other |
| <ol> <li>The PI certifies that if this individual will conduct any clinical activities as part of this study, the individual is appropriately credentialed and privileged to practice within the institution where the research will be conducted: Individual has no clinical responsibilities</li> </ol> |
| 6. * Qualifications to carry out study related responsibilities: (you may select multiple answers) |
| Education and/or Professional Preparation |
| Experience - Research |
| Experience - Clinical |
| Experience - Related Skills |

| HM20024502 |
|------------|

7. Additional or Emergency Phone:

View: SF - Community Engaged Research HM20024502 ID: HM20024502

# Community Engaged Research

If this pop-out window fails to respond after you click OK, close the window and email the responses you were trying to enter here to ERAHelp@vcu.edu. This pop-out window has a known system glitch. ERA Help personnel can assist with entering this information for you.

- 1. \* Name of the organization: Islamic center of Richmond
- 2. \* Zip code or country of the organization: 23060
- 3. \* Select the role that best describes this community partner/co-researchers:

- Provides guidance to the researcher about the study design, subject recruitment, data collection, or data analysis. Partner/Co-researcher does NOT make decisions about study design.
- Makes decisions WITH the researcher about the study's research activities and/or helps conduct those activities (i.e., study design, subject recruitment, data collection, and/or data analysis)

139/155

HM20024502 7/8/23, 9:07 AM

HM20024502

ID: HM20024502

View: SF\_IRB\_Summary\_Document

## Add Document

1. \* Document Name: Consent form focus group

2. \* Type: Consent/Assent/Information Sheet

3. \* File:

Namoos- Consent from of focus group 05.12.2023.pdf(0.03)

HM20024502 7/8/23, 9:07 AM

HM20024502 ID: HM20024502

View: SF\_IRB\_Summary\_Document

## Add Document

1. \* Document Name: Consent form - Intervention program

2. \* Type: Consent/Assent/Information Sheet

3. \* File:

☑ Namoos- Consent from of Intervention group 05.12.2023 copy.pdf(0.04)

HM20024502 7/8/23, 9:07 AM

HM20024502

ID: HM20024502

View: SF\_IRB\_Summary\_Document

## Add Document

1. \* Document Name: Fund Plan

2. \* Type: Funding Proposal

3. \* File:

Asmaa -Budget 04.13.2023.xlsx(0.03)

View: SF\_IRB\_Summary\_Document HM20024502 ID: HM20024502 7/8/23, 9:07 AM

## Add Document

1. \* Document Name: Education session

**2. \* Type:** Other

3. \* File:

Asmaa Education session guide , intervention group- 04.07.2023.docx(0.02)
View: SF\_IRB\_Summary\_Document HM20024502 ID: HM20024502

# Add Document

1. \* Document Name: Timeline Plan

**2. \* Type:** Other

3, \* File:

HM20024502 ID: HM20024502

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: Conceptual model

2. \* Type: Research Measure

3. \* File:

Asmaa Conceptual Model 05.12.2023.docx(0.02)

ID: HM20024502

7/8/23, 9:07 AM

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: Flayer 2

**2. \* Type:** Other

3. \* File:

型劃 Asmaa Flyer Version 05.12.2023.docx(0.01)

HM20024502

ID: HM20024502

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: Namoos-Focus group script guide

**2. \* Type:** Other

3. \* File:

Namoos -Focus Group Script Guide.docx(0.02)

HM20024502

View: SF\_IRB\_Summary\_Document

HM20024502 Add Document ID: HM20024502

1. \* Document Name: Participants -RA communication script

**2. \* Type:** Other

3, \* File:

Mamoos- Participants -RA communication script .docx(0.01)

HM20024502

ID: HM20024502

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: Study Survey( Pre-post and satisfactory scales)

2. \* Type: Research Measure

3, \* File:

Survey- Promise women project 05.12.2023.docx(0.01)

HM20024502

ID: HM20024502

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: consent form- focus group

2. \* Type: Consent/Assent/Information Sheet

3, \* File:

(0.01) Consent from -Focus group 02.20.2023.docx

HM20024502 ID: HM20024502

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: VS biosketch

2. \* Type: CV/Biosketch

3, \* File:

Sheppard Biosketch for AN 11.14.2022.pdf(0.01)

HM20024502

ID: HM20024502

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: Communication log

**2. \* Type:** Other

3. \* File:

Communication log.docx(0.01)

HM20024502

ID: HM20024502

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: PRMC approval

2. \* Type: Ancillary Committee Approval

3. \* File:

2022-10-10\_MCC-22-19873\_PRMC Approval Letter.pdf(0.01)

HM20024502

ID: HM20024502

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: Flyer

**2. \* Type:** Other

3, \* File:

Hyer 004.08.2022.png(0.01)

HM20024502

ID: HM20024502

View: SF\_IRB\_Summary\_Document

# Add Document

1. \* Document Name: Namoos Resume

2. \* Type: CV/Biosketch

3, \* File:

Dr. Namoos A. Biosketch 06.07.2021.pdf(0.01)